Evaluation of Toric Soft Contact Lenses Containing a Chromophore to Block High-Energy Visible Light Produced on Commercial Manufacturing Lines

Protocol CR-6484

Version: 1.0

Date: 14 March 2022

Investigational Products: Test lens: Rotationally stabilized astigmatic contact lens in senofilcon A (C3) with a chromophore to block High-Energy Visible Light (HEVL), control lens: ACUVUE® OASYS® 1-Day for Astigmatism

Keywords: Astigmatism, toric contact lenses, senofilcon A (C3), RTY-1 chromophore, HEVL, dispensing, daily wear, daily disposable, visual acuity, CLUE Comfort, CLUE Vision, CLUE Handling, logMAR visual acuity, rotation performance, cosmetic acceptability, ACUVUE® OASYS® 1-Day for Astigmatism, Single use Eye-Cept® Rewetting Drops, LacriPure Saline Solution, ScleralFil Preservative Free Saline Solution.

#### Statement of Compliance to protocol, GCP and applicable regulatory guidelines:

This trial will be conducted in compliance with the protocol, ISO 14155:2020,<sup>1</sup> the International Council for Harmonization Good Clinical Practice E6(R2) (ICH GCP),<sup>2</sup> the Declaration of Helsinki,<sup>3</sup> and all applicable regulatory requirements.

#### **Confidentiality Statement:**

This document contains confidential information, which should not be copied, referred to, released or published without written approval from Johnson & Johnson Vision Care, Inc. The information may not be disclosed to others except to the extent necessary to obtain Institutional Review Board/Independent Ethics Committee approval and informed consent, or as required by International, Federal and State Laws, as applicable. Persons to whom this information is disclosed must be informed that this information is privileged and confidential and that it should not be further disclosed without the written permission of Johnson & Johnson Vision Care, Inc. Any supplemental information that may be added to this document is also confidential and proprietary to Johnson & Johnson Vision Care, Inc. and must be kept in confidence in the same manner as the contents of this document.

| | E OF CONTENTS<br>DCOL TITLE, NUMBER, VERSION AND DATE | 6 |
|---|---|---|
| | SOR NAME AND ADDRESS | |
| | CAL MONITOR | _ |
| | ORIZED SIGNATURES | |
| | GE HISTORY | |
| | PSIS | |
| | IONLY USED ABBREVIATIONS, ACRONYMS AND DEFINITION | |
| 1. IN | TRODUCTION AND BACKGROUND | 16 |
| 1.1. | Name and Descriptions of Investigational Products | 16 |
| 1.2. | Intended Use of Investigational Products | 16 |
| 1.3. | Summary of Findings from Nonclinical Studies | 16 |
| 1.4. | Summary of Known Risks and Benefits to Human Subjects | 16 |
| 1.5.<br>Study | Relevant Literature References and Prior Clinical Data Relevant to Pr<br>y 17 | oposed Clinical |
| 2. ST | TUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES | 17 |
| 2.1. | Objectives | 17 |
| 2.2. | Endpoints | 17 |
| 2.3. | Hypotheses | 18 |
| 3. TA | ARGETED STUDY POPULATION | 18 |
| 3.1. | General Characteristics | 18 |
| 3.2. | Inclusion Criteria | 18 |
| 3.3. | Exclusion Criteria | 19 |
| 3.4. | Enrollment Strategy | 20 |
| 4. ST | TUDY DESIGN AND RATIONALE | 20 |
| 4.1. | Description of Study Design | 20 |
| 4.2. | Study Design Rationale | 20 |
| 4.3. | Enrollment Target and Study Duration | 21 |
| 5. TE | EST ARTICLE ALLOCATION AND MASKING | 21 |
| 5.1. | Test Article Allocation | 21 |
| 5.2. | Masking | 22 |
| 5.3. | Procedures for Maintaining and Breaking the Masking | 22 |
| 6 ST | TIDY INTERVENTION | 22 |

| | 6.1. | Identity of Test Articles | 22 |
|----|-------|--------------------------------------------------|----|
| | 6.2. | Ancillary Supplies/Products | 23 |
| | 6.3. | Administration of Test Articles | 24 |
| | 6.4. | Packaging and Labeling | 24 |
| | 6.5. | Storage Conditions | 24 |
| | 6.6. | Collection and Storage of Samples | 25 |
| | 6.7. | Accountability of Test Articles | 25 |
| 7. | STU | UDY EVALUATIONS | 26 |
| | 7.1. | Time and Event Schedule | 26 |
| | 7.2. | Detailed Study Procedures | 27 |
| | VIS | SIT 1 | 27 |
| | VIS | SIT 2 | 33 |
| | VIS | SIT 3 | 35 |
| | VIS | SIT 4 | 36 |
| | FIN | IAL EVALUATION | 37 |
| | 7.3. | Unscheduled Visits | 38 |
| | 7.4. | Laboratory Procedures | 39 |
| 8. | SU | BJECTS COMPLETION/WITHDRAWAL | 39 |
| | 8.1. | Completion Criteria. | 39 |
| | 8.2. | Withdrawal/Discontinuation from the Study | 40 |
| 9. | PR | E-STUDY AND CONCOMITANT INTERVENTION/MEDICATION | 40 |
| | 9.1. | Systemic Medications | 40 |
| 1( | ). D | EVIATIONS FROM THE PROTOCOL | 42 |
| 1 | 1. S' | TUDY TERMINATION | 43 |
| 12 | 2. P | ROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS | 44 |
| 1. | 3. A | DVERSE EVENTS | 45 |
| | 13.1. | Definitions and Classifications | 45 |
| | 13.2. | Assessing Adverse Events | 47 |
| | 13. | 2.1. Causality Assessment | 47 |
| | 13. | 2.2. Severity Assessment | 48 |
| | 13.3. | Documentation and Follow-Up of Adverse Events | 48 |
| | 13.4. | Reporting Adverse Events | 49 |
| | 13.4 | 4.1. Reporting Adverse Events to Sponsor | 50 |

| | 13.4. | 2. Reporting Adverse Events to the Responsible IEC/IRB and Health Auth 50 | oritie |
|---|---|---|---|
| 13 | 3.5. | Event of Special Interest | 51 |
| 13 | 3.6. | Reporting of Pregnancy | 51 |
| 14. | ST | ATISTICAL METHODS | 51 |
| 14 | <b>l</b> .1. | General Considerations | 51 |
| 14 | 1.2. | Sample Size Justification | 51 |
| 14 | 1.3. | Analysis Populations | 52 |
| 14 | 1.4. | Level of Statistical Significance | 53 |
| 14 | 1.5. | Primary Analysis | 53 |
| 14 | 1.6. | Secondary Analysis | 53 |
| 14 | 1.7. | Other Exploratory Analysis | 53 |
| 14 | 1.8. | Interim Analysis | 54 |
| 14 | 1.9. | Procedure for Handling Missing Data and Drop-Outs | 54 |
| 14 | 1.10. | Procedure for Reporting Deviations from Statistical Plan | 54 |
| 15. | DA | TA HANDLING AND RECORD KEEPING/ARCHIVING | |
| 15 | 5.1. | Electronic Case Report Form/Data Collection | 54 |
| 15 | 5.2. | Subject Record | 55 |
| 15 | 5.3. | Trial Registration on ClinicalTrials.gov | 55 |
| 16. | DA | TA MANAGEMENT | 55 |
| 16 | 5.1. | Access to Source Data/Document | 55 |
| 16 | 5.2. | Confidentiality of Information. | 55 |
| 16 | 5.3. | Data Quality Assurance | 56 |
| 16 | 5.4. | Data Monitoring Committee (DMC) | 56 |
| 17. | CL | INICAL MONITORING | 56 |
| 18. | ET | HICAL AND REGULATORY ASPECTS | 57 |
| 18 | 3.1. | Study-Specific Design Considerations | 57 |
| 18 | 3.2. | Investigator Responsibility | 57 |
| 18 | 3.3. | Independent Ethics Committee or Institutional Review Board (IEC/IRB) | 57 |
| 18 | 3.4. | Informed Consent | 58 |
| 18 | 3.5. | Privacy of Personal Data | 59 |
| 19. | ST | UDY RECORD RETENTION | 60 |
| 20. | FIN | NANCIAL CONSIDERATIONS | 60 |
| 21 | ΡIJ | BLICATION | 61 |

| 22. REFERENCES | 61 |
|---|---|
| APPENDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES) | 62 |
| APPENDIX B: PATIENT INSTRUCTION GUIDE | 78 |
| APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT) | 79 |
| APPENDIX D: | 108 |
| LENS FITTING CHARACTERISTICS | |
| SUBJECT REPORTED OCULAR SYMPTOMS | 115 |
| DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACT | |
| BIOMICROSCOPY SCALE | 123 |
| DISTANCE AND NEAR VISUAL ACUITY EVALUATION | 129 |
| TORIC FIT EVALUATION | 134 |
| ETDRS DISTANCE VISUAL ACUITY MEASURMENT PROCEDURE | 139 |
| PATIENT REPORTED OUTCOMES | 143 |
| LENS INSERTION AND REMOVAL | 145 |
| VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINA TESTING | |
| APPENDIX E: IRIS COLOR SCALE | 157 |
| APPENDIX F: GUIDELINES FOR COVID-19 RISK MITIGATION | 158 |
| PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE | 170 |
| LIST OF TABLES Table 1: Ancillary Supplies | 24 |
| Table 2: Time and Events | |
| Table 3: Disallowed systemic medications | |
| Table 4: Disallowed systemic antihistamines | |
| Table 5: Examples of major and minor protocol deviations | |
| Table 6: Power Calculation for the Primary Hypothesis of CLUE Comfort score inferiority of the Test relative to the Control) with Type I error of 0.05 | • |
| LIST OF FIGURES | |
| Figure 1: Study Flowchart | 14 |

#### PROTOCOL TITLE, NUMBER, VERSION AND DATE

Title: Evaluation of Toric Soft Contact Lenses Containing a Chromophore to Block High-

Energy Visible Light Produced on Commercial Manufacturing Lines

Protocol Number: CR-6484

Version: 1.0

Date: 14 March 2022

#### SPONSOR NAME AND ADDRESS

Johnson & Johnson Vision Care, Inc. (JJVC) 7500 Centurion Parkway Jacksonville, FL 32256

#### **MEDICAL MONITOR**



The Medical Monitor must be notified by the clinical institution/site by e-mail or telephone within 24 hours of learning of a Serious Adverse Event. The Medical Monitor may be contacted during business hours for adverse event questions. General study related questions should be directed towards your assigned clinical research associate.

The Medical Monitoring Plan is maintained as a separate document and included in the Trial Master File.

#### **AUTHORIZED SIGNATURES**

The signatures below constitutes the approval of this protocol and the attachments and provide the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable U.S. federal regulations,<sup>4</sup> ISO 14155:2020,<sup>1</sup> ICH guidelines,<sup>2</sup> and the Declaration of Helsinki.<sup>3</sup>

| Author & Study<br>Responsible Clinician | See Electronic Signature Report | |
|---|---|---|
| Clinical Operations | | DATE |
| Manager | See Electronic Signature Report | DATE |
| Biostatistician | See Electronic Signature Report | DATE |
| Data Management | See Electronic Signature Report | DATE |
| Medical Safety<br>Officer | See Electronic Signature Report | DATE |
| Approver | See Electronic Signature Report | DATE |

#### **CHANGE HISTORY**

| Version | Originator | Description of Change(s) and | Justification for | Date |
|---|---|---|---|---|
| | | Section Number(s) Affected | Change | |
| 1.0 | | Original Protocol | N/A | 14 Mar 2022 |

#### **SYNOPSIS**

| Protocol Title | Evaluation of Toric Soft Contact Lenses Containing a Chromophore to Block High-Energy Visible Light Produced |
|---|---|
| | on Commercial Manufacturing Lines |
| Sponsor | JJVC, 7500 Centurion Parkway, Jacksonville, FL 32256 |
| Clinical Phase | Clinical trial phase: Confirmatory |
| | Design control phase: Development phase, phase 2b |
| Trial Registration | This study will be registered on ClinicalTrials.gov by the Sponsor. |
| Test Article(s) | Investigational Products: Test lens: Rotationally stabilized |
| | astigmatic soft contact lens in senofilcon A (C3) with a |
| | chromophore to block High-Energy Visible Light (HEVL). |
| | Approved Products: Control lens: ACUVUE® OASYS® |
| | 1-Day for Astigmatism (AO1DfA) |
| Wear and Replacement | Wear Schedule: Daily wear |
| Schedules | Replacement Schedule: Daily disposable |
| Objectives | Primary Objective: |
| | The primary objective of this study is to evaluate and compare |
| | the subjective CLUE Comfort score for the test lens against the control lens. The following hypothesis will be tested: |
| | • The test lens is non-inferior to the control lens with |
| | respect to overall CLUE Comfort score at follow-up. |
| | A non-inferiority margin of -5 points on the CLUE |
| | scale will be used. |
| | Exploratory Objectives: |
| | Exploratory objectives of this study will be to evaluate the |
| | subjective CLUE Vision, subjective CLUE Handling, lens |
| | fitting characteristics, rotational performance, visual acuity, |
| | ocular physiological response and cosmetic acceptability for |
| | the test and control designs. |

| Study Endpoints | Primary endpoints: |
|---|---|
| | <ul> <li>Responses to the CLUE questionnaire Comfort items<br/>at the follow-up visit</li> </ul> |
| | Other observations: |
| | HLHC distance VA at the follow-up visit |
| | • Lens fitting characteristics (centration, movement, and |
| | push-up test) at dispensing and follow-up visits |
| | <ul> <li>Settled lens orientation at the dispensing visit and at<br/>follow-up visits</li> </ul> |
| | Lens rotational stability with blinks at the dispensing visit |
| | Subjective response to MRD questionnaire items at the follow-up visit |
| | Subjective response to the CLUE questionnaire Comfort, Vision and Handling items at fitting |
| | Subjective response to the CLUE questionnaire Vision and Handling items at follow-up |
| | Slit lamp findings across all study visits |
| | Adverse events |
| Study Design | This will be a 4-visit, randomized, controlled, single-masked, |
| | bilateral wear, dispensing, 2-treament, 2-sequence, 3-period |
| | crossover study. Each subject will be randomized into one of |
| | two unique sequences to wear two different study lenses one |
| | at a time over three wear periods (test/control/control or |
| | control/test/test). During each wear period the lenses will be |
| | worn bilaterally for approximately 1 week (7±2 days) in a |
| | daily disposable modality. Subjective CLUE Comfort, Vision and Handling will be assessed using the CLUE questionnaire |
| | at both fitting and follow-up visits for each wear period. |
| | HLHC VA will be assessed at the follow-up evaluation using |
| | ETDRS charts. There will be no washout period between wear |
| | periods. |
| | See the flow chart at the end of the synopsis table for the |
| | schematic of the study visits and procedures of main |
| G 1 G' | observations (Figure 1). |
| Sample Size | This study will have an enrollment target of approximately |
| | 140 subjects, with a target of at least 126 to complete (assuming a dropout rate of 10%). |
| Study Duration | Total study duration including the enrollment period is |
| Stady Dalation | anticipated to be approximately 10 weeks. |
| Anticipated Study | Subjects will be habitual bilateral soft contact lens wearers |
| Population | with bilateral astigmatism who are between 18 and 39 years |
| | of age (inclusive). |

| Eligibility Criteria - | Potential subjects must satisfy of all the following criteria to |
|---|---|
| Inclusion | be enrolled in the study. |
| | Inclusion Criteria following Screening |
| | The subject must: |
| | 1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form. |
| | 2. Appear able and willing to adhere to the instructions set forth in this clinical protocol. |
| | 3. Be between 18 and 39 years of age (inclusive) at the time of screening. |
| | 4. Habitually wear soft contact lenses in both eyes in a daily or daily disposable wear modality (i.e., not extended wear modality). Habitual wearer is defined as a minimum of 6 hours per day, for a minimum of 2 days per week during the past four weeks. |
| | 5. Possess a wearable pair of spectacles that provide correction for distance vision. |
| | Inclusion Criteria at Baseline Evaluation |
| | The subject must: |
| | 6. In both eyes, have refractive error suitable for correction |
| | with the toric contact lens powers available in this study: a. Sphere powers (DS) -1.50 through -4.00 in 0.25 steps b. Cylinder powers (DC) -0.75 and -1.25 |
| | c. Axes (°) 170, 180, 10, 80, 90, 100 |
| | 7. Have best corrected monocular distance visual acuity of 20/30 or better in each eye. |

## Eligibility Criteria – Exclusion

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

Exclusion Criteria following Screening

The subject must not:

- 1. Be currently pregnant or lactating.
- 2. Be diabetic.
- 3. Be currently using any ocular medications or have an ocular infection of any type.
- 4. By self-report, have any ocular or systemic disease, allergies, infection, or use of medication that might contraindicate or interfere with contact lens wear, or otherwise compromise study endpoints, including (e.g., infectious disease hepatitis. tuberculosis). contagious immunosuppressive disease (e.g., Human Immunodeficiency Virus [HIV]), autoimmune disease (e.g. rheumatoid arthritis, Sjögren's syndrome), or history of serious mental illness or seizures. See section 9.1 for additional details regarding excluded systemic medications.
- 5. Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (e.g. SynergEyes, SoftPerm) within the past 6 months.
- 6. Be currently wearing monovision or multifocal contact lenses.
- 7. Be currently wearing lenses in an extended wear modality.
- 8. Have a history of strabismus or amblyopia.
- 9. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site.
- 10. Have participated in a contact lens or lens care product clinical trial within 7 days prior to study enrollment.

Exclusion Criteria following Baseline Evaluation The subject must not:

11. Have clinically significant (grade 3 or higher on the FDA grading scale) slit lamp findings (e.g., corneal edema, neovascularization or staining, tarsal abnormalities or bulbar injection) or other corneal or ocular disease or abnormalities that contraindicate contact lens wear or may otherwise compromise study endpoints (including entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis).

| | <ul> <li>12. Have fluctuations in vision due to clinically significant dry eye or other ocular conditions.</li> <li>13. Have had or have planned (within the study period) any ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, iridotomy, retinal laser photocoagulation, etc.).</li> </ul> |
|---|---|
| Disallowed | Subjects will not be eligible to enroll if they are taking any |
| Medications/Interventions | ocular medications, or any systemic medications that would<br>normally contraindicate contact lens wear or may otherwise<br>compromise study endpoints. See section 9.1 for details<br>regarding disallowed systemic medications. |
| Measurements and Procedures | Key procedures associated with the endpoints for this study will include: |
| | <ul> <li>Overseeing completion of subjective questionnaires</li> <li>Measurement of HLHC VA using ETDRS charts at follow-up</li> </ul> |
| | - Examination of the anterior segment using a slit lamp biomicroscope and grading findings using the FDA grading scale |
| | - Assessment of general lens fitting characteristics (centration, movement, push-up test) |
| | - Assessment of lens orientation and rotational stability using a slit lamp biomicroscope |
| Microbiology or Other Laboratory Testing | Not applicable for this study. |
| Study Termination | The occurrence of an Unanticipated Adverse Device Effect (UADE) or Serious Adverse Event (SAE) for which a causal relationship to a test article cannot be ruled out, will result in stopping further dispensing investigational product. In the event of a UADE or SAE, the Sponsor Medical Monitor may unmask the treatment regimen of subject(s) and may discuss this with the Principal Investigator before any further subjects are enrolled. |
| Ancillary Supplies/ Study- | Lens cases, fluorescein strips and preservative-free rewetting |
| Specific Materials | drops / artificial tears will be supplied for use as needed. |
| Principal Investigator(s) | A full list of Principal Investigators, clinical sites, and |
| and Study | institutions is kept separately from the Study Protocol and is |
| Institution(s)/Site(s) | included in the study Trial Master File. |

Figure 1: Study Flowchart



## COMMONLY USED ABBREVIATIONS, ACRONYMS AND DEFINITIONS OF TERMS

ADE Adverse Device Effect

ADHD Attention Deficit Hyperactivity Disorder
AE Adverse Event/Adverse Experience

AO1DfA ACUVUE OASYS® 1-DAY with HydraLuxe<sup>TM</sup> TECHNOLOGY for

**ASTIGMATISM** 

BSCVA Best Spectacle Corrected Visual Acuity

CFR Code of Federal Regulations
CLUE Contact Lens User Experience
COM Clinical Operations Manager
CRA Clinical Research Associate

CRF Case Report Form

CRO Contract Research Organization

D Diopter

DMC Data Monitoring Committee
eCRF Electronic Case Report Form
EDC Electronic Data Capture
ESD Eyelid Stabilized Design

ETDRS Early Treatment Diabetic Retinopathy Study

FDA Food and Drug Administration

GCP Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act

HIV Human Immunodeficiency Virus

IB Investigator's Brochure

ICH The International Council for Harmonization

IEC Independent Ethics Committee IRB Institutional Review Board

ISO International Organization for Standardization

ITT Intent-to-Treat

JJVC Johnson & Johnson Vision Care, Inc.

LASIK Laser-Assisted in Situ Keratomileusis

LogMAR Logarithm of Minimal Angle of Resolution

OD Right Eye
OS Left Eye
OU Both Eyes

PIG Patient Instruction Guide
PQC Product Quality Complaint
PRK Photorefractive Keratectomy
PRO Patient Reported Outcome

OA Quality Assurance

SAE Serious Adverse Event/Serious Adverse Experience

SAS Statistical Analysis System

SD Standard Deviation

UADE Unanticipated Adverse Device Effect

USADE Unanticipated Serious Adverse Device Effect

VA Visual Acuity

#### 1. INTRODUCTION AND BACKGROUND

High Energy Visible Light (HEVL) may be generally defined as the visible region of the electromagnetic spectrum with wavelengths shorter than 500 nm. Due to Rayleigh scattering, light within this range of wavelengths is scattered more than light of longer wavelengths, thus filtering these shorter wavelengths may result in increased visual contrast when looking at distant objects. At approximately 435 nm, visible light has enough energy to damage the retinal pigment epithelium and has been linked to macular degeneration. Additionally, the retinal receptors responsible for photoentrainment (entrainment of the circadian rhythm in response to patterns of light and dark) are maximally sensitive to light at approximately 480 nm.

Ophthalmic lenses that block High Energy Visible Light (HEVL) may offer improved vision through enhanced chromatic contrast sensitivity. Such lenses may also provide greater retinal protection than regular lenses without spectral filtering. This study will investigate the subjective visual response to a daily disposable, toric lens design incorporating a HEVL-blocking chromophore (RTY-1) against the ACUVUE® OASYS 1-Day for ASTIGMATISM (AO1DfA) design as control.

#### 1.1. Name and Descriptions of Investigational Products

The test lens in this study will be a toric contact lens design with stabilization design and geometry similar to AO1DfA in senofilcon A (C3) with the addition of a HEVL-blocking chromophore (RTY-1). The test lens will be evaluated against the AO1DfA lens in as control.

Further details about the test and control articles are given in section 6 of this protocol.

#### 1.2. Intended Use of Investigational Products

The intended use of the investigational products is the correction of myopic astigmatism. Study lenses will be worn bilaterally in a daily wear, daily disposable modality for at least 8 hours per day and 5 days per week over a wear period of 7±2 days. Three wear periods will be completed in total, with no washout period between the wear periods.

#### 1.3. Summary of Findings from Nonclinical Studies

All previous pre-clinical findings were deemed satisfactory prior to proceeding with clinical trials on humans. For the most comprehensive nonclinical information regarding the test and control designs refer to the latest version of the Investigator's Brochure<sup>5</sup> and the AO1DfA package insert (Appendix C), respectively.

#### 1.4. Summary of Known Risks and Benefits to Human Subjects

The anticipated clinical benefit of the investigational lenses will be the correction of refractive error. No adverse device effects are anticipated. The risks associated with use of the

investigational lenses are considered to be the same as those for other marketed soft contact lens worn in the same modality (i.e., daily disposable wear). No additional risks associated with participation in this investigation are anticipated.

Comprehensive risk and benefit information regarding the test design and the AO1DfA control lens are included in the latest versions of the Investigator's Brochure<sup>5</sup> and the AO1DfA package insert (Appendix C), respectively.

## 1.5. Relevant Literature References and Prior Clinical Data Relevant to Proposed Clinical Study



In study , out of the 98 subjects included in the safety population, one ocular adverse event (AE) was reported; non-significant meibomianitis was reported in the right eye of one subject, and this was considered to have no relation to the investigational articles or study procedures. No ocular adverse events were reported in.

In study \_\_\_\_\_\_, 144 subjects were included in the safety population and no ocular adverse events were reported throughout the study period.

For further details regarding literature references and prior clinical data related to the test designs and the AO1DfA control lens, refer to the Investigator's Brochure<sup>5</sup> and the AO1DfA package insert (Appendix C), respectively.

#### 2. STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES

#### 2.1. Objectives

Primary Objective

The primary objective of this study is to evaluate and compare the subjective CLUE Comfort of the HEVL-blocking test design against AO1DfA as control.

#### **Exploratory Objectives**

Exploratory objectives of this study will be to evaluate the subjective CLUE Vision, subjective CLUE Handling, lens fitting characteristics, rotation performance, visual acuity, ocular physiological response and cosmetic acceptability for the test and control designs.

#### 2.2. Endpoints

Primary Endpoint

The primary endpoint will be the responses to the CLUE questionnaire Comfort items at the follow-up evaluation.

Subjective comfort will be assessed using Contact Lens User Experience (CLUE) questionnaire. CLUE is a validated patient-reported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses (Comfort, Vision, Handling, and Packaging) in a contact-lens wearing population in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response. A 5-point increase in an average CLUE score translates into 10% shift in the distribution of scores for population of soft disposable contact lens wearers.

The CLUE questionnaire was selected for the primary endpoint since this is thought to be the best psychometric method available for evaluating and quantifying subjective lens comfort. The follow-up CLUE questionnaire was selected since this allows the ample time for subjects to subjectively assess lens performance over a variety of wear conditions.

Other Exploratory Endpoints

- HLHC distance VA at the follow-up visit
- Lens fitting characteristics (centration, movement, and push-up test) at dispensing and follow-up visits
- Settled lens orientation at the dispensing visit and at follow-up visits
- Lens rotational stability with blinks at the dispensing visit
- Subjective response to MRD questionnaire items at the follow-up visit
- Subjective response to the CLUE questionnaire Comfort, Vision, and Handling items at fitting
- Subjective response to the CLUE questionnaire Vision and Handling items at followup
- Slit lamp findings across all study visits
- Adverse events

#### 2.3. Hypotheses

Primary Hypothesis

The following hypothesis will be tested:

• The test lens is non-inferior to the control with regard to the CLUE Comfort score at the follow-up evaluation. A non-inferiority margin of -5 CLUE points will be used.

#### 3. TARGETED STUDY POPULATION

#### 3.1. General Characteristics

The target population for this study will be healthy adult soft contact lens wearers between 18 and 39 years of age with binocular myopic astigmatism.

#### 3.2. Inclusion Criteria

Potential subjects must satisfy of all the following criteria to be enrolled in the study.

Inclusion Criteria following Screening

#### The subject must:

- 1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
- 2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
- 3. Be between 18 and 39 years of age (inclusive) at the time of screening.
- 4. By self-report, habitually wear soft contact lenses in both eyes in a daily or daily disposable wear modality (i.e. not extended wear modality). Habitual wearer is defined as a minimum of 6 hours per day, for a minimum of 2 days per week during the past four weeks.
- 5. Possess a wearable pair of spectacles that provide correction for distance vision.

#### Inclusion Criteria at Baseline Evaluation

#### The subject must:

- 6. In both eyes, have refractive error suitable for correction with the toric contact lens powers available in this study:
  - a. Sphere powers (DS) -1.50 through -4.00 in 0.25 steps
  - b. Cylinder powers (DC) -0.75 and -1.25
  - c. Axes (°) 170, 180, 10, 80, 90, 100
- 7. Have best corrected monocular distance visual acuity of 20/30 or better in each eye.

#### 3.3. Exclusion Criteria

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

#### Exclusion Criteria following Screening

The subject must not:

- 1. Be currently pregnant or lactating.
- 2. Be diabetic.
- 3. Be currently using any ocular medications or have an ocular infection of any type.
- 4. By self-report, have any ocular or systemic disease, allergies, infection, or use of medication that might contraindicate or interfere with contact lens wear, or otherwise compromise study endpoints, including infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive disease (e.g., Human Immunodeficiency Virus [HIV]), autoimmune disease (e.g. rheumatoid arthritis, Sjögren's syndrome), or history of serious mental illness or seizures. See section 9.1 for additional details regarding excluded systemic medications.
- 5. Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (e.g. SynergEyes, SoftPerm) within the past 6 months.
- 6. Be currently wearing monovision or multifocal contact lenses.
- 7. Be currently wearing lenses in an extended wear modality.
- 8. Have a history of strabismus or amblyopia.
- 9. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site.
- 10. Have participated in a contact lens or lens care product clinical trial within 7 days prior to study enrollment.

Exclusion Criteria at Baseline Evaluation

The subject must not:

- 11. Have clinically significant (grade 3 or higher on the FDA grading scale) slit lamp findings (e.g., corneal edema, neovascularization or staining, tarsal abnormalities or bulbar injection) or other corneal or ocular disease or abnormalities that contraindicate contact lens wear or may otherwise compromise study endpoints (including entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis).
- 12. Have fluctuations in vision due to clinically significant dry eye or other ocular conditions.
- 13. Have had or have planned (within the study period) any ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, iridotomy, retinal laser photocoagulation, etc.).

#### 3.4. Enrollment Strategy

Study subjects will be recruited from the Institution/clinical site's subject database and/or utilizing Independent Ethics Committee (IEC) or Institutional Review Board (IRB) approved materials.

#### 4. STUDY DESIGN AND RATIONALE

#### 4.1. Description of Study Design

This will be a 4-visit, randomized, controlled, single-masked, bilateral wear, dispensing, 2-treatment, 2-sequence, 3-period crossover study. Each subject will be randomized into one of two unique sequences to wear two different study lenses one at a time over three wear periods (test/control/control or control/test/test). During each wear period, study lenses will be worn bilaterally for approximately 1 week (7±2 days) in a daily disposable modality. Study lenses will be worn for a minimum of 8 hours per day and at least 5 days per week during each wear period. Subjective CLUE Comfort, Vision and Handling will be assessed using the CLUE questionnaire at both fitting and follow-up visits for each wear period. HLHC VA will be assessed at the follow-up evaluation using ETDRS charts. There will be no washout period between wear periods. Subjects will not have access to the study lenses following completion of the protocol.

#### 4.2. Study Design Rationale

A crossover study design was chosen to allow each subject to act as their own active control. A 3-period design was chosen to allow estimation of first-order carryover effects.

The AO1DfA lens was chosen as control since this is thought to be the best performing currently marketed ACUVUE® toric lens in terms of comfort. The prescribed wear schedule (lenses to be worn for a minimum of 8 hours per day and a minimum of 5 days per week) was chosen as this is representative of a typical wear schedule for contact lens wearers.

For the primary study endpoint, the CLUE questionnaire was selected on the basis of being the best available validated PRO tool for assessing the subjective comfort of soft contact lens wearers.

The investigational lenses will be fitted by optometrists who are experienced at fitting toric soft contact lenses and will be evaluated by habitual contact lens wearers in their standard wearing environment.

#### 4.3. Enrollment Target and Study Duration

This study will have an enrollment target of 140 subjects, with a target of at least 126 to complete. The study will be conducted at up to 12 clinical sites, where the enrollment target for each site will be approximately 10 to 20 subjects. A subject will be considered enrolled upon signing of the informed consent form.

There will be 4 visits in total per subject; total study duration including the enrollment period is expected to be approximately 10 weeks. The investigation will end with completion of the final subject's last visit. Subjects who are discontinued prior to the final evaluation may be replaced at the discretion of the study sponsor. The investigation will end at the time that the study data is hard locked.

#### 5. TEST ARTICLE ALLOCATION AND MASKING

#### 5.1. Test Article Allocation

This study will be a randomized, single-masked, crossover design. Subjects will be randomized into one of two unique sequence groups in a 1:1 allocation ratio to wear two different study lens designs (test and control designs) one at a time bilaterally over three wear periods.

Use of the test articles will be randomized using a randomization scheme supplied by the study biostatistician. The randomized assignment of subjects will be performed at the first visit prior to the first fitting. Clinical sites will follow the randomization scheme provided and will not pre-select or assign subjects. The following must have occurred prior to randomization:

- Informed consent must have been obtained
- The subject must have met all inclusion and exclusion criteria
- The subject history and baseline information must have been collected

Randomly permuted block randomization will be used to avoid bias in the assignment of subjects to treatment and to enhance the validity of statistical comparisons across treatment groups.

When dispensing test articles, the following steps should be followed to maintain randomization codes:

1. Investigator or designee (documented on the Delegation Log) will consult the randomization scheme (lens fitting schedule) to obtain the test article assignment for that subject prior to dispensing.

- 2. Investigator or designee will record the subject's number on the appropriate line of the randomization scheme (lens fitting schedule).
- 3. Investigator or designee will pull the appropriate test articles from the study supply. All test articles that are opened, whether dispensed (placed/fit on eye or dispensed outside the clinical site) or not, must be recorded on the Test Article Accountability Log in the "Dispensed" section.

#### 5.2. Masking

To reduce the potential for bias, this will be a single-masked trial; subjects will not be aware of the identity of the assigned lenses, however, due to the difference in appearance of the test lenses containing the RTY-1 chromophore, it is expected that subjects will be able to visually differentiate between the test and control designs. The identity (i.e., brand and type) of the study lenses will be masked by having the blister packs labeled with the study number, lot number, sphere power, cylinder power, axis, expiration date and randomization code. Investigators, site staff and sponsor personnel (including the medical monitor) will be aware of the identity of the test and control lenses.

#### 5.3. Procedures for Maintaining and Breaking the Masking

Under normal circumstances, the mask should not be broken until all subjects have completed the study and the database is finalized. Otherwise, the mask should be broken only if specific emergency treatment/course of action would be dictated by the subject knowing their treatment status. In such cases, the Investigator may, in an emergency, contact the medical monitor. In the event the mask is broken, the Sponsor must be informed as soon as possible. The date, time, and reason for the unmasking must be documented in the subject record.

Subjects who have had their treatment assignment unmasked are expected to return for all remaining scheduled evaluations. Subjects who are discontinued may be replaced at the discretion of the study sponsor.

#### 6. STUDY INTERVENTION

#### **6.1.** Identity of Test Articles

The following contact lenses will be used in this study:

| | Test | Control |
|---|---|---|
| Test Article Form | Soft contact lens | |
| | TRA100 and TRA200 series | AO1DfA |
| Design / Description | toric contact lens with HEVL- | |
| | blocking chromophore | |
| Design Name | | AO1DfA |
| Manufacturer | Johnson & Johnson Vision Care, Inc. | |
| Packaging Form | Blister packaging in sterile packing solution | |
| Packaging Solution | Optimized Borate Buffer (OBB) solution | |

| Lens Material | senofilcon A (C3) with RTY-1<br>chromophore | senofilcon A (C3) |
|---|---|---|
| Sphere Powers (DS) | -1.50 to -4.00 in 0.25 steps | |
| Cylinder Powers (DC) | -0.75, -1.25 | |
| Cylinder Axes (°) | 10, 80, 90, 1 | 00, 170, 180 |
| Nominal Water<br>Content (%) | 4 | 1 |
| Nominal Base<br>Curve (mm) | 8. | .5 |
| Lens Diameter (mm) | 14.3 | |
| Fiducial marks | 6 and 12 o'clock fiducial lines | |
| Dk (Fatt method,<br>boundary corrected,<br>edge corrected, ×10 <sup>-11</sup> [cm <sup>2</sup> /sec] [ml<br>O <sub>2</sub> /ml × mm Hg] at<br>35°C) | 103 | |
| Modality in Current<br>Study | Daily wear | |
| Replacement Frequency in Current Study | Daily disposable | |

In total, both test and control lenses will be available in 132 unique lens powers (11 sphere powers  $\times$  2 cylinder powers  $\times$  6 axes).

For each study lens design (test and control), the total number of test lenses to be used in this study (not including lenses that are replaced due to droppage, loss or damage) is expected to be approximately 2940 lenses (target enrollment of 70 subjects × 2 eyes per subject × 7 days per wear period × 2 wear periods for the first sequence, plus 70 subjects × 2 eyes per subject × 7 days per wear period × 1 wear period for the second sequence).

#### 6.2. Ancillary Supplies/Products

The following solutions will be used in this study:

Table 1: Ancillary Supplies

| | Non-Preserved Rewetting Drops | | |
|---|---|---|---|
| | Single use Eye- | LacriPure Saline | ScleralFil |
| Solution Name/Description | Cept® Rewetting | Solution | Preservative Free |
| | Drops | | Saline Solution |
| Manufacturer | Optics Laboratory | Menicon | Bausch & Lomb |
| Preservative | None | None | None |

Lens cases and fluorescein strips (either 0.6 mg or 1.0 mg) will be supplied for use as needed.

#### 6.3. Administration of Test Articles

Test articles will be dispensed to subjects meeting all eligibility requirements, including any dispensing requirements set forth in this clinical protocol. Subjects will be dispensed an adequate supply of test articles to complete the study. Lost or damaged test articles may be replaced at the discretion of the investigator and/or the sponsor.

#### 6.4. Packaging and Labeling

The test articles will be supplied in blister packages as the primary packaging and placed into plastic bags as secondary packaging. Test and control blister packages will be physically overlabeled with permanent labels. Representative sample labels for the primary and secondary packaging are shown below:



#### **6.5.** Storage Conditions

Test articles will be maintained at ambient temperatures at the clinical site. Test articles must be kept under secure conditions.

#### 6.6. Collection and Storage of Samples

No samples will be collected as part of the study procedures. When possible, any lens or test article associated with an Adverse Event and/or a Product Quality Complaint must be retained and stored in a glass vial with moderate solution pending directions from the sponsor for potential return to JJVC.

#### 6.7. Accountability of Test Articles

JJVC will provide the Investigator with sufficient quantities of study articles and supplies to complete the investigation. The Investigator is asked to retain all lens shipment documentation for the test article accountability records.

Test articles must be kept in a locked storage cabinet, accessible only to those assigned by the Investigator for dispensing. The Investigator may delegate this activity to authorized study site personnel listed on the Site Delegation Log. All test articles must be accounted. This includes:

- 1. What was dispensed for the subject for trial fitting, to wear out of the office, or issued for the subject to replace appropriately between visits.
- 2. What was returned to the Investigator unused, including expired or malfunctioning product.
- 3. The number and reason for unplanned replacements.

The Investigator will collect all unused test articles from the subjects at the end of the subject's participation. Subject returned unused test articles must be separated from the clinical study inventory of un-dispensed test articles and must be labeled with the subject number and date of return. Following final reconciliation of test articles by the monitor, the Investigator or monitor will return all unused test articles to JJVC.

If there is a discrepancy between the shipment documents and the contents, contact the study monitor <u>immediately</u>.

#### 7. STUDY EVALUATIONS

#### 7.1. Time and Event Schedule

Table 2: Time and Events

| Visit Information | Visit 1 Screening, Baseline, Lens Fitting #1 | Visit 2 Follow-up #1, Lens Fitting #2 | Visit 3 Follow-up #2, Lens Fitting #3 | Visit 4 Follow-up #3, Final Evaluation |
|---|---|---|---|---|
| Time Point | Day 0 | 7 ± 2 days<br>following<br>Visit 2 | 7 ± 2 days<br>following<br>Visit 3 | 7 ± 2 days<br>following<br>Visit 4 |
| Minimum lens wear time immediately prior to visit | Must wear habitual lenses | 1 hour (study lenses) | 1 hour (study lenses) | 1 hour (study lenses) |
| Estimated Visit Duration | 2.5 hours | 2.5 hours | 2.5 hours | 1.5 hours |
| Statement of informed consent | X | | | |
| Demographics | X | | | |
| Medical history/concomitant medications | X | X | X | X |
| Habitual contact lens information | X | | | |
| Habitual lens wear time | X | | | |
| Eligibility at Screening | X | | | |
| Subject reported ocular symptoms | X | X | X | X |
| Baseline PRO questionnaire | X | | | |
| Entrance visual acuity | X | X | X | X |
| Remove habitual lenses | X | | | |
| Subjective Sphero-Cylindrical Refraction | X | | | X |
| Slit Lamp Biomicroscopy | X | X | X | X |
| Eligibility at Baseline | X | | | |
| Iris color | X | | | |
| Lens Selection | X | X | X | |
| Lens insertion and timed rotation assessments | X | X | X | |
| Lens settling | X | X | X | |
| Toric fit assessment | X | X | X | |
| General fit assessment | X | X | X | |
| Spherical over-refraction | X | X | X | |
| Lens modification (if necessary) | X | X | X | |
| Post-fit PRO questionnaire | X | X | X | |
| Additional samples of toric lens orientation (performed twice) | Х | х | х | х |
| Exit visual acuity | X | X | X | |
| Dispensing criteria | X | X | X | |
| Dispensing instructions | X | X | X | |

| Visit Information | Visit 1 Screening, Baseline, Lens Fitting #1 | Visit 2 Follow-up #1, Lens Fitting #2 | Visit 3<br>Follow-up<br>#2, Lens<br>Fitting #3 | Visit 4 Follow-up #3, Final Evaluation |
|---|---|---|---|---|
| Time Point | Day 0 | 7 ± 2 days<br>following<br>Visit 2 | 7 ± 2 days<br>following<br>Visit 3 | 7 ± 2 days<br>following<br>Visit 4 |
| Minimum lens wear time immediately prior to visit | Must wear habitual lenses | 1 hour (study lenses) | 1 hour (study lenses) | 1 hour (study lenses) |
| Estimated Visit Duration | 2.5 hours | 2.5 hours | 2.5 hours | 1.5 hours |
| Schedule next visit | X | X | X | |
| Wear time and compliance | | X | X | X |
| Collect unworn lenses | | X | X | X |
| Follow-up PRO questionnaire | | X | X | X |
| Distance HLHC visual acuity using ETDRS charts | | X | X | X |
| Toric lens orientation | | X | X | X |
| Lens removal | | X | X | X |
| Continuance | | X | X | |
| Subject completion status | | | | X |

#### 7.2. Detailed Study Procedures

#### VISIT 1

Subjects must wear their habitual contact lenses to this visit.

| | Visit 1: Screening | |
|---|---|---|
| Step | Procedure | Details |
| 1.1 | Statement of Informed | Each subject must read, understand, and sign the |
| | Consent | Statement of Informed Consent before being |
| | | enrolled into the study. The Principal Investigator |
| | | or his/her designee conducting the informed |
| | | consent discussion must also sign the consent |
| | | form. |
| | | <b>Note:</b> The subject must be provided a signed |
| | | copy of this document. |
| 1.2 | Demographics | Record the subject's year of birth, age, gender, |
| | | race and ethnicity. |
| 1.3 | Medical History and | Record the subject's medical history and |
| | Concomitant | concomitant medications. |
| | Medications | |

| | Visit 1: Screening | |
|---|---|---|
| Step | Procedure | Details |
| 1.4 | Habitual Lenses | Record the subject's habitual lens type, parameters, lens care solution, wear modality and approximate prescription date. |
| 1.5 | Habitual lens wear time. | Record the average and comfortable wear time for the subject's habitual contact lenses. |
| 1.6 | Eligibility after<br>Screening | All responses to Screening Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria must be answered "no" for the subject to be considered eligible. If subject is deemed to be ineligible after screening, proceed to Final Evaluation and complete Subject Disposition. Refraction and Biomicroscopy forms do not need to be completed as part of Final Evaluation. |

| | | Visit 1: Baseline |
|---|---|---|
| Step | Procedure | Details |
| 1.7 | Subject reported ocular symptoms | Record any subject reported ocular symptoms reported with regard to their habitual contact lenses. |
| 1.8 | Baseline PRO questionnaire | Ask the subject to fill out the baseline questionnaire regarding their experience with their <b>habitual contact lenses</b> . |
| 1.9 | Entrance visual acuity | Record the monocular distance Snellen visual acuity for each eye (OD, OS) to the nearest letter with the subject's habitual contact lens correction. Subjects must continue until at least 50% of the letters on a line are read incorrectly. |
| 1.10 | Remove habitual lenses | The subject's habitual contact lenses will be removed and stored in a lens case, if required. |
| 1.11 | Subjective sphero-<br>cylindrical refraction | Conduct a full spherocylindrical bare eye subjective refraction with binocular balance and record the resultant monocular visual acuity for each eye to the nearest letter. Note: The duo-chrome test should be used for |
| | | refining the monocular and binocular spherical endpoints. This test will be considered to have reached the endpoint when the targets on red and green backgrounds appear to be equally sharp. |
| | | However, if the subject's response changes immediately from "red" to "green" with a 0.25DS change in power, the endpoint will be the most plus power (with "red" target clearer) before this reversal. |

| | Visit 1: Baseline | |
|---|---|---|
| Step | Procedure | Details |
| 1.12 | Slit lamp<br>biomicroscopy | The FDA Slit Lamp Classification Scale will be used to grade findings. If any slit lamp finding is graded as 3 or worse, the visit will be discontinued; however, the subject may repeat the baseline evaluation (one time) at a later date once the condition lessens. |
| | | Should the clearance of the fluorescein need to be expedited, preservative free rewetting drops or artificial tears may be instilled. |
| 1.13 | Eligibility at baseline | All responses to Inclusion Criteria questions must<br>be answered "yes" and all responses to Exclusion<br>Criteria questions must be answered "no" for the<br>subject to be considered eligible. |
| | | If subject is deemed to be ineligible after baseline, proceed to Final Evaluation. |
| 1.14 | Iris color | The investigator will record the subject's iris color using the scale provided (Appendix E). |

| Visit 1: Lens Fitting #1 | | |
|---|---|---|
| Step | Procedure | Details |
| 1.15 | Lens selection | Assign the study lens based on the randomization scheme. Select the fitting lens powers based on vertex-corrected subjective refraction for each eye, with consideration of the following guidelines: |
| | | <ol> <li>Label cylinder axis should be determined by rounding the refraction cylinder axis to the nearest 10 degrees. Axis ending in the digit '5' should be rounded towards 180 for eyes with with-the-rule astigmatism, or towards 90 for eyes with against-the-rule astigmatism (e.g. 175 should be rounded to 180, 105 should be rounded to 100).</li> <li>Cylinder power should be chosen based on the following table:</li> </ol> |
| | | Vertex corrected cylinder power (X) within the range: (DC) Label cylinder power to be fit (DC) |
| | | $-0.625 \le X < -1.125$ $-0.75$ |
| | | $-1.125 \le X < -1.625$ $-1.25$ |
| | | 3. The fitting lens spherical equivalent (SE) power (label sphere power + 1/2 of the label |

| | Visit 1: Lens Fitting #1 | |
|---|---|---|
| Step | Procedure | Details |
| | | cylinder power) should be as close as possible to the SE of the vertex-corrected refraction. If the SE of the vertex-corrected refraction is exactly halfway between two label SE powers, the least minus label power should be fit first. |
| 1.16 | Right eye lens insertion | Instruct the subject to insert the right-eye lens with random orientation. If lens is uncomfortable, inspect for damage and |
| 1.17 | Timed rotation<br>assessments during<br>settling period | remove, reinsert or replace as necessary. Start a stopwatch (or suitable smartphone or tablet timing app) as soon as the right lens is inserted. Record lens rotation (direction and magnitude) to the nearest degree at one (1) and three (3) minutes following insertion. |
| | | Note: All lenses in this study have scribe marks at 6 o'clock and 12 o'clock positions and rotation measurements are made relative to a vertical reference line. |
| 1.18 | Left eye lens insertion | Instruct the subject to insert the left-eye lens with random orientation. If lens is uncomfortable, inspect for damage and remove, reinsert or replace as necessary. |
| 1.19 | Timed rotation<br>assessments during<br>settling period | Start a stopwatch (or suitable smartphone or tablet timing app) as soon as the left lens is inserted. Record lens rotation (direction and magnitude) to the nearest degree at one (1) and three (3) minutes following insertion. Note: All lenses in this study have scribe marks at 6 o'clock and 12 o'clock positions and rotation measurements are made relative to a vertical reference line. |
| 1.20 | Lens settling | Allow lenses to settle for a period of at least 10 minutes following left lens insertion. |

| | | Visit 1: Lens Fitting #1 |
|---|---|---|
| Step | Procedure | Details |
| 1.01 | T | D 10 1 |
| 1.21 | Toric fit assessment | Record for each eye: 1. The rotational position to the nearest degree 2. Lens stability with blinks 3. Toric fit acceptability. The toric lens fit will be designated as 'unacceptable' if either: |
| | | a. The lens ABSOLUTE ROTATION is greater than 20 degrees b. The LENS STABILITY WITH BLINK is greater than 5 degrees If one or both lenses demonstrate an unacceptable toric fit, the subject will be discontinued (proceed to final evaluation). |
| 1.22 | General lens fit assessment | The fitting characteristics of the lens in both eyes will be assessed using a slit lamp. Lens position (centration, limbal exposure, edge lift) and movement (primary and up gaze as well as pushup) will be assessed. Fit acceptability is defined as any lens that does <b>not</b> display the following general fit characteristics: <ul> <li>Limbal exposure (presence of clear cornea) in any direction of gaze.</li> <li>Edge lift</li> <li>Insufficient movement in all three movement assessments (primary gaze, upgaze and push-up test).</li> <li>Excessive movement in primary gaze</li> </ul> If the general fit is unacceptable for either eye, the subject will be discontinued (proceed to exit evaluation). |
| 1.23 | Spherical over-refraction | Perform monocular spherical over-refraction using duo-chrome to refine the endpoint as described in step 1.11 (the final spherical endpoint may be determined binocularly). The spherical over-refraction must be plano in both eyes to continue. If a non-plano over-refraction is found in either eye, the lens(es) must be refit with the indicated change in sphere power. If the indicated lens power is not available for either eye (e.g., outside the available SKU range), the subject will be discontinued (proceed to final evaluation). |

| | Visit 1: Lens Fitting #1 | |
|---|---|---|
| Step | Procedure | Details |
| 1.24 | Lens modification (if necessary) | If modification is necessary in one or both eyes, select the reason for refitting lenses: • The settled lens rotation is such that a different cylinder axis would be more appropriate (use the LARS rule to determine the replacement lens cylinder axis) • The spherical over-refraction is not plano • Other (specify reason) Repeat steps 1.16 through 1.23 for one or both eyes, as appropriate. A maximum of 2 lens modifications are allowed per eye. If, for either eye, the fit is not successful after 2 modifications, the subject will be discontinued (proceed to final evaluation). |
| 1.25 | Post-fit PRO questionnaire | Subjects will complete a PRO questionnaire regarding the initial comfort, vision and handling of the study lenses. |
| 1.26 | Additional sample of toric lens orientation (1) | Instruct the subject to leave the consulting room and walk around for at least 2 minutes. Upon their return, measure and record the toric lens orientation for each eye to the nearest degree. |
| 1.27 | Additional sample of toric lens orientation (2) | Repeat the previous step once again. |
| 1.28 | Exit visual acuity | Record the exit monocular distance Snellen visual acuity for each eye with the subject wearing the study lenses. |
| 1.29 | Dispensing criteria | Lenses may be dispensed if both following conditions are met: 1. The monocular distance visual acuity with the study lenses is equal to or better than 20/25 in each eye. 2. The subject indicates that the comfort and vision with the study lenses is acceptable. If either of these conditions is not met, the subject will be discontinued (proceed to exit evaluation). |
| 1.30 | Dispensing instructions | <ul> <li>If the study lenses are suitable for dispensing:</li> <li>Instruct the subject to wear the study lenses for at least 8 hours per day (in a daily wear / daily disposable modality) on at least 5 days of the wear period. Subjects must not wear their habitual lenses at any time during the dispensing period.</li> </ul> |

| | Visit 1: Lens Fitting #1 | |
|---|---|---|
| Step | Procedure | Details |
| | | Provide the subject with a copy of the Patient Instruction Guide. |
| | | Preservative-free rewetting drops are permitted, if needed. |
| | | Dispense enough lenses for the subject to complete the wear period (i.e. up to and including their scheduled follow-up visit). At the investigator's discretion, in instances where there is a high likelihood of the subject needing replacement lenses (e.g., due to subject activities, unavailability of subject or site during the wear period, high likelihood of lens tears, etc.), one additional spare pair may be dispensed. |
| | | Note: In the event that a subject requires additional lenses due to loss or damage, they may return to the clinical site for lens replacement. As much as reasonably possible, damaged lenses and packaging should be returned to the clinical site (in solution, if possible) for shipping to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form, store the lens in a labeled vial with saline and return it to the Sponsor. |
| | | Ensure the subject is aware of the correct lens power for each eye (label the lenses with R and L as appropriate). |
| 1.31 | Schedule next visit | Schedule the follow-up visit to occur in $7 \pm 2$ days (counting the day of this visit as day 0, the subject may return on day 5 through 9). Ensure the subject is instructed to wear the study lenses for at least 1 hour immediately prior to attending the follow-up visit. |

#### VISIT 2

Visit 2 will occur 5 to 9 days following Visit 1. Subjects must present to this visit wearing the study lenses in both eyes, and lenses must have been worn for at least 1 hour prior to the visit.

| Visit 2: Follow-Up #1 | | | | | |
|---|---|---|---|---|---|
| Step | Procedure | Details | | | |
| 2.1 | Wear time and compliance | Record the subjects wearing time and comfortable wearing time. Subjects must have worn lenses for at least five 8-hour (continuous) periods during the dispensing period, and for at least 1 hour prior to attending this visit. | | | |
| 2.2 | Collect unworn lenses | Collect any unworn study lenses that were dispensed at the previous visit. | | | |
| 2.3 | Review medical<br>history and<br>concomitant<br>medications | Record any changes to the subject's medical history (including adverse events) or concomitant medications. | | | |
| 2.4 | Subject reported ocular symptoms | Record any subject reported ocular symptoms in response to a verbal open-ended symptoms questionnaire. | | | |
| 2.5 | Follow-up PRO questionnaire | Subjects will complete a PRO questionnaire to assess their experience with the study lenses. Note: at the end of the second wear period (Visit 3: Follow-Up #2) the PRO questionnaire will also include questions regarding lens preference between the lenses worn in the first and second wear periods. | | | |
| 2.6 | Entrance visual acuity | Record the entrance Snellen VA for each eye while wearing the study lenses. | | | |
| 2.7 | Distance ETDRS visual acuity | Measure monocular distance high luminance high contrast (HLHC) visual acuity using ETDRS charts at 4 meters. | | | |
| Measure each eye using the charts table below: | | | | | he |
| | | Condition | HL | НС | |
| | | Room illumination > 400 lux | | 0 lux | |
| | | Chart luminance | 120 - 20 | 00 cd/m <sup>2</sup> | |
| | | Eye | OD | OS | |
| | | Charts | HC-1<br>HC-2 | HC-3<br>HC-4 | |
| 2.6 | | Recorded letter-by-lett | | | |
| 2.8 | Toric lens orientation | Record the toric lens orientation for each eye to the nearest degree. | | | |
| 2.9 | Additional sample of toric lens orientation (1) | Instruct the subject to leave the consulting room and walk around for at least 2 minutes. Upon their return, measure and record the toric lens orientation to the nearest degree in each eye. | | | |

| Visit 2: Follow-Up #1 | | |
|---|---|---|
| Step | Procedure | Details |
| 2.10 | Additional sample of toric lens orientation (2) | Repeat the previous step once again. |
| 2.11 | Lens removal | Remove and place both lenses into a lens case with saline solution. |
| | | Do not discard the lenses until after biomicroscopy has been completed. |
| 2.12 | Biomicroscopy | The FDA Slit Lamp Classification Scale will be used to grade findings. If any slit lamp finding is graded as 3 or worse, the subject must be discontinued, an adverse event will be recorded, and the subject will be monitored as per the guidelines given in section 13. Should the clearance of the fluorescein need to be expedited, preservative free rewetting drops or artificial tears may be instilled. Study lenses may be discarded if there is no reason to store them following biomicroscopy. |
| 2.13 | Continuance | Verify that the subject is eligible to continue with the study. |

#### Visit 2: Lens Fitting #2

The steps followed will be the same as those listed under Visit 1: Lens Fitting #1.

#### VISIT 3

Visit 3 will occur 5 to 9 days following Visit 2. Subjects must present to this visit wearing the study lenses in both eyes, and lenses must have been worn for at least 1 hour prior to the visit.

The steps followed will be the same as those listed under Visit 2: Follow-Up #1, with the addition of a Preference Questionnaire as part of the Follow-Up PRO questionnaire step.

### Visit 3: Lens Fitting #3

The steps followed will be the same as those listed under Visit 1: Lens Fitting #1.

#### VISIT 4

Visit 4 will occur 5 to 9 days following Visit 3. Subjects must present to this visit wearing the study lenses in both eyes, and lenses must have been worn for at least 1 hour prior to the visit. Subjects should bring their own habitual spectacles or contact lenses to this visit to wear following study lens removal.

| Visit 4: Follow-Up #3 | | | | | | | |
|---|---|---|---|---|---|--|--|
| Step | Procedure | Details | | | | | |
| 4.1 | Wear time and compliance | Record the subjects wearing time and comfortable wearing time. Subjects must have worn lenses for at least five 8-hour (continuous) periods during the dispensing period, and for at least 1 hour prior to attending this visit. | | | | | |
| 4.2 | Collect unworn lenses | Collect any unworn study lenses that were dispensed at the previous visit. | | | | | |
| 4.3 | Review medical history and concomitant medications | Record any changes to the subject's medical history (including adverse events) or concomitant medications. | | | | | |
| 4.4 | Subject reported ocular symptoms | Record any subject reported ocular symptoms in response to a verbal open-ended symptoms questionnaire. | | | | | |
| 4.5 | Follow-up PRO questionnaire | Subjects will complete a PRO questionnaire to assess their experience with the study lenses. | | | | | |
| 4.6 | Entrance visual acuity | Record the entrance Snellen VA for each eye while wearing the study lenses. | | | | | |
| 4.7 | Distance ETDRS visual acuity | Measure monocular distance high luminance high contrast (HLHC) visual acuity using ETDRS charts at 4 meters. | | | | | |
| | | Measure each eye using below: | ble | | | | |
| | | Condition | HLHC | | ] | | |
| | | Room illumination | > 40 | 0 lux | | | |
| | | Chart luminance | 120 - 200 cd/m <sup>2</sup> | | ] | | |
| | | Eye | OD | OS | ] | | |
| | | Charts | HC-1 | HC-3 | 1 | | |
| | | | HC-2 | HC-4 | | | |
| | | Recorded letter-by-letter results into EDC. | | | | | |
| 4.8 | Toric lens orientation | Record the toric lens orientation for each eye to the nearest degree. | | | | | |
| | Visit 4: Follow-Up #3 | | | |
|---|---|---|--|--|
| Step | Procedure | Details | | |
| 4.9 | Additional sample of toric lens orientation (1) | Instruct the subject to leave the consulting room and walk around for at least 2 minutes. Upon their return, measure and record the toric lens orientation to the nearest degree in each eye. | | |
| 4.10 | Additional sample of toric lens orientation (2) | Repeat the previous step once again. | | |
| 4.11 | Lens removal | Remove and place both lenses into a lens case with saline solution. | | |
| | | Do not discard the lenses until after biomicroscopy has been completed. | | |
| 4.12 | Biomicroscopy | The FDA Slit Lamp Classification Scale will be used to grade findings. If any slit lamp finding is graded as 3 or worse, an adverse event will be recorded, and the subject will be monitored as per the guidelines given in section 13. Should the clearance of the fluorescein need to be expedited, preservative free rewetting drops or artificial tears may be instilled. | | |
| | | Study lenses may be discarded if there is no reason to store them following biomicroscopy. | | |

## FINAL EVALUATION

The final evaluation will ordinarily take place immediately following the last scheduled follow-up visit per the study protocol. It may also take place at any point the subject discontinues the study or is terminated from the study.

| | Final Evaluation | |
|---|---|---|
| Step | Step Procedure Details | |
| F.1 | Final Exam Form | Indicate if the subject completed the study |
| | (subject completion | successfully. If subject discontinued from the |
| | status) | study, indicate the reason. |
| F.2 Exit Refraction Perform bare-eye subjective spherocylindrical refraction with a phoropter and record the best-corrected distance visual acuity (OD and OS) to the nearest letter. | | |
| | Note: This step is not necessary if the subject was exited due to screen failure. | |

| | Final Evaluation | |
|---|---|---|
| Step | Step Procedure Details | |
| F.3 | Exit Slit Lamp Biomicroscopy (for subjects that are | FDA Slit Lamp Classification Scale will be used to grade the findings. |
| | discontinued early) | If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. This step is not necessary if the subject was exited due to screen failure. |
| | | <b>Note</b> : This step is not necessary if the subject was exited due to screen failure, or if biomicroscopy was performed as part of the final follow-up visit procedures (i.e., immediately prior to the final evaluation). |

#### 7.3. Unscheduled Visits

If, during the investigation, a subject requires an unscheduled visit to the clinical site, the following information will be collected, as appropriate:

- Chief complaint prompting the visit. If the reason is an adverse event, the applicable eCRF for the adverse event must be completed and subject record completed as appropriate.
- Date and time of the visit and all procedures completed at the unscheduled visit.
- Review of adverse event and concomitant medications.
- Documentation of any test article dispensed or collected from the subject, if applicable.
- Slit lamp findings (using the Slit Lamp Classification Scale).

If the Investigator withdraws a subject from the study, the final study visit case report forms must be completed indicating the reason(s) why the subject was withdrawn. The subject record must be completed documenting the date and primary reason for withdrawal and the study CRA notified.

Any ocular and non-ocular Adverse Events that are ongoing at the time of the study visit will be followed by the Investigator, within licensure, until they have resolved, returned to pretreatment status, stabilized, or been satisfactorily explained. If further treatment i.e., beyond licensure is required, the subject will be referred to the appropriate health care provider.

The following information will be collected during an unscheduled visit.

| | Unscheduled Visit | |
|---|---|---|
| Step | Procedure | Details |
| U.1 | Reason for | Indicate if the <u>only</u> reason for the visit is that the |
| | unscheduled visit subject requires additional test articles. If the | |
| | | reason is other than resupply of previously |
| | | dispensed lenses, specify the reason for the visit. |
| U.2 | Chief Complaints (if | Record the subject's chief complaints for reasons |
| | applicable) | for the unscheduled visit. |

| | Unscheduled Visit | |
|---|---|---|
| Step | Procedure | Details |
| U.3 | Adverse Events and<br>Concomitant<br>Medications Review<br>(if applicable) | Review any changes to the subject's medical history or concomitant medications from the previous study visit. Record any changes, and any adverse events. |
| U.4 | Entrance VA (if applicable) | Record the entrance distance visual acuity (OD, OS) to the nearest letter. |
| U.5 | Subjective Spherocylindrical Refraction (if applicable) | Perform bare-eye subjective spherocylindrical refraction with a phoropter (adopt the maximum plus to maximum visual acuity (MPMVA) approach and use the duo-chrome test for binocular balancing) and record the best corrected distance visual acuity to the nearest letter (OD, OS). |
| U.6 | Slit Lamp<br>Biomicroscopy (if<br>applicable) | FDA Slit Lamp Classification Scale will be used to grade the findings. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. |
| U.7 | Dispensing (if applicable) | If the subject requires additional lenses to complete the wear period and is eligible to do so, provide additional lenses per the dispensing instructions given in the detailed study procedures. |
| U.8 | Exit Visual Acuity (if applicable) | Record the subject's exit distance visual acuity (OD, OS) to the nearest letter. |

NOTE: If the only reason for the unscheduled visit is that the subject requires additional test articles, only the dispensing information needs to be recorded.

# 7.4. Laboratory Procedures

Not applicable.

### 8. SUBJECTS COMPLETION/WITHDRAWAL

## 8.1. Completion Criteria

Subjects are considered to have completed the study if they:

- provided informed consent.
- they are eligible.
- have not withdrawn/discontinued from the study for any reason described in section 8.2.
- completed all visits through the final visit (visit 4). If all visits were completed but an additional visit is considered necessary for subject care, follow the requirements for unscheduled visits in section 7.3.

### 8.2. Withdrawal/Discontinuation from the Study

A subject will be withdrawn from the study for any of the following reasons:

- Subject withdrawal of consent.
- Subject not compliant to protocol.
- Subject lost to follow-up.
- Subject no longer meets eligibility criteria (e.g. the subject becomes pregnant).
- Subject develops significant or serious adverse events necessitating discontinuation of study lens wear.
- Subjects who have experienced a Corneal Infiltrative Event (CIE).
- Investigator's clinical judgment regarding the subject safety reasons (that it is in the best interest of the subject to stop treatment).
- Subject misses any study visits.
- Subject not compliant with study lens wear schedule.
- Subject not successfully dispensed due to lack of efficacy and safety including poor vision, poor comfort, or unacceptable fit.

For discontinued subjects, the Investigator will:

- Complete the current visit (scheduled or unscheduled).
- Complete the Final Evaluation, indicating the reason that the subject was discontinued from the study.
- Record the spherocylindrical refraction with best corrected distance visual acuity.
- Collect used test article(s) (worn or brought to the visit) from the subject and discard them, unless otherwise stated in section 7.2.
- Collect all unused test article(s) from the subject.
- Make arrangements for subject care, if needed, due to their study participation

Additional subjects may be enrolled if a subject discontinues from the study prematurely.

In cases where a subject is lost to follow-up, every possible effort must be made to contact the subject and determine the reason for discontinuation/withdrawal. The measures taken to follow up must be documented including two written attempts and a certified letter (or equivalent) as the final attempt.

#### 9. PRE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION

Concomitant medications will be documented during screening and updated during the study. Disallowed concomitant interventions for this study include ocular medications of any kind, or any systemic medications that would normally contraindicate contact lens wear or may otherwise compromise study endpoints.

# 9.1. Systemic Medications

Certain systemic medications are known to have a higher likelihood to interfere with contact lens wear, chiefly by disrupting the tear film.

A summary of disallowed systemic medications is shown in Table 3. Subjects with a history of taking these medications will be allowed to enroll only if:

- The medications have been taken on a continual, routine basis for at least 6 months, and
- The subject has demonstrated successful contact lens wear during this time.

Or:

• The subject was taking the medication on a temporary basis and ceased taking that medication at least 2 weeks prior to signing the informed consent (this is considered sufficient time for the medication to have left the body prior to enrollment).

Subjects with a history of taking medications listed in Table 3 on a long-term, routine basis for less than 6 months will not be allowed to participate in the study.

Table 3: Disallowed systemic medications

| Class of Drug | Common Indication(s) | Common Examples |
|---|---|---|
| Estrogens (not including contraceptive medication) | Menopause, osteoporosis, vaginitis | Vagifem, Estrace, Climara, Vivelle-Dot, Premarin, Minivelle, etc. |
| Anticholinergics | Irritable bowel syndrome,<br>Parkinson's disease, peptic ulcer,<br>cystitis, nasal congestion, cold<br>symptoms, overactive bladder,<br>COPD | Symax SL, Homax SL, Cogentin, |
| Beta-blockers | Hypertension, angina, heart attack, migraine, artrial fibrillation, andrenal cancer, essential tumor, glaucoma | Toprol XL, Lopressor, Tenormin, Propranolol, Timoptic, Trandate, Inderal LA, etc. |
| Psychotropics | Antipsychotic (schizophrenia, mania), antidepression, antiobsessive, antianxiety, mood stabilizer, stimulants (ADHD) | Zoloft, Celexa, Prozac, Lexapro,<br>Effexor, Cymbalta, Ativan,<br>Xanax, Desyrel, Wellbutrin, etc. |
| Vitamin A<br>analogs | Cystic acne | Isotretinoin |

Examples of disallowed systemic antihistamines are given in Table 4. Subjects with a history of taking systemic antihistamines will be allowed to enroll only if:

- They have taken antihistamines continuously for at least 2 weeks, and
- They have demonstrated successful wear while taking the medication

Or:

• They stopped taking the medication for at least 2 weeks prior to enrollment.

Table 4: Disallowed systemic antihistamines

| Class of Drug | Common Indication(s) | Common Examples |
|----------------|----------------------|-----------------|
| Antihistamines | | |

#### 10. DEVIATIONS FROM THE PROTOCOL

Investigator will notify study sponsor upon identification of a protocol deviation. Protocol deviations must be reported to the sponsor within 24 hours after discovery of the protocol deviation. The Investigator will report deviations per IRB/IEC requirements. All deviations will be tracked, and corrective actions implemented as appropriate.

If it becomes necessary for the Investigator to implement a deviation in order to eliminate an immediate hazard to the trial subject, the Investigator may implement the deviation immediately without notification to the sponsor. Within 24 hours after the implemented deviation, the Investigator must notify and provide the rationale to the Sponsor and, as required, the IEC/IRB.

If the deviation potentially impacts the safety of patient or changes the technical integrity of the study, then it must be reported to IEC/IRB. This is a "Major Deviation". Deviations that contradict the information contained in the Informed Consent/Assent forms will be considered Major Deviations.

Minor deviations have no substantive effect on patient safety or technical integrity of the study. They are often logistical in nature.

Protocol waivers are prohibited.

Table 5 lists examples of deviations that will constitute major and minor protocol deviations for this study.

Table 5: Examples of major and minor protocol deviations

| <b>Deviation category</b> | Major deviation | Minor deviation |
|---|---|---|
| Out-of-window visit | • | Visit attended ≤ 2 days out of visit window defined in study procedures. |
| Unanswered PRO questions | For questionnaires where data is related to a primary endpoint, more than 2 PRO | data is related to a primary or |

| <b>Deviation category</b> | Major deviation | Minor deviation |
|---|---|---|
| | questions are unanswered (i.e., left blank). | fewer PRO questions are unanswered (i.e., left blank). |
| | For questionnaires not related to the primary endpoint, the questionnaire is not completed (i.e., all questions are unanswered). | |
| Insufficient wear of study lenses | Subject does not wear study lenses for at least 8 hours on at least 5 days of a study lens wear period. | Subject does not wear study lenses for at least 1 hour prior to attending a follow-up visit. |
| | Subject wears their habitual lenses during any of the study lens wear periods. | |

In the case of a major protocol deviation, the decision of whether or not the subject will be excluded from the Per-Protocol analysis population will be made at the time of cohort review.

#### 11. STUDY TERMINATION

The occurrence of one or more Unanticipated Serious Adverse Device Effect (USADE), or any SAE where the relationship to study agent cannot be ruled out, may result in stopping further dispensing of test article. In the event of a USADE or SAE, the Sponsor may unmask the treatment regimen for the subject(s) and will discuss this with the Investigator before any further subjects are enrolled.

The Sponsor will determine when a study will be stopped. The Principal Investigator always has the discretion to initiate stopping the study based on patient safety or if information indicates the study's results are compromised.

JJVC reserves the right to terminate the study at any time for any reason. Additionally, the IEC/IRB reserves the right to terminate the study if an unreasonable risk is determined. The study can be terminated by the Principal Investigator at the individual clinical site due to specific clinical observations, if in their opinion, after a discussion with JJVC, it is determined that it would be unwise to continue at the clinical site.

JJVC (and the IEC/IRB and DMC, if applicable) will evaluate all adverse events. If it is determined that an adverse event presents an unreasonable risk, the investigation, or that part of the investigation presenting the risk, will be terminated as soon as possible.

Should the study be terminated (either prematurely or as scheduled), the Investigator will notify the IEC/IRB and Regulatory Authority as required by local regulatory requirements.

## 12. PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS

A Product Quality Complaint (PQC) refers to any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness or performance of test articles after they have been released for clinical trial use.

Potential complaints may come from a variety of sources including but not limited to subjects, clinical research associates (CRA), clinical operations managers (COM), medical monitors, and site personnel, etc. The following are not considered product quality complaints:

- Subject satisfaction inquiries reported via "Subjective Questionnaires" and "Patient Reported Outcomes (PRO)."
- Clinical test articles that are stored improperly or damaged after receipt at the investigational site.
- Lens replacements that occur due to drops/fall-outs.
- Damage deemed by clinicians or clinical staff to be caused by handling by the user, and not indicative of a quality deficiency (i.e. tears, rips, etc.), only in situations where there is no deficiency alleged by the subject.

Within 24 hours of site personnel becoming aware that a PQC has occurred, the PQC must be recorded in the EDC system, which will trigger an automatic email notification to the appropriate COM/CRA and Clinical QA representative. In cases where the EDC system in use is not configured to send automatic notifications or when an EDC system is not used, the COM/CRA is responsible for notifying Clinical QA upon discovery that a PQC has occurred.

Upon receipt of the EDC notification, the COM/CRA will contact the study site to collect additional information which will include:

- Date the complaint was received/recorded in the EDC System (Date of Sponsor Awareness).
- Who received the complaint.
- Study number.
- Clinical site information (contact name, site ID, telephone number).
- Lot number(s).
- Unique Subject Identifier(s).
- Indication of who first observed complaint (site personnel or subject).
- OD/OS indication, along with whether the lens was inserted.
- Any related AE number if applicable.
- Detailed complaint description (scheduled/unscheduled visit, wear time, symptoms, resolution of symptoms, etc.).
- Eye Care Provider objective (slit lamp) findings if applicable.

• Confirmation of product availability for return (and tracking information, if available), or rationale if product is not available for return

Once a complaint is received, it will be assessed by the COM, CRA, or trained site personnel to determine if it is an Adverse Event/Serious Adverse Event (AE/SAE). If the complaint results in an AE/SAE, the COM/CRA, or trained site personnel will follow section 13 of this protocol. If the AE/SAE was potentially the result of a product quality related deficiency, these procedures also applies and will be executed in parallel.

In some cases, a PQC form may be generated in EDC by the site in error. In this event, the PQC forms will be marked "Intentionally Left Blank" or "ILB". Justification for ILB must be documented.

#### 13. ADVERSE EVENTS

#### 13.1. Definitions and Classifications

**Adverse Event (AE)** – An AE is "any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device."

**Note**: This definition includes events related to the investigational medical device or the comparator, and to the procedures involved. For users or other persons, this definition is restricted to events related to investigational medical devices.<sup>1</sup>

An AE includes any condition (including a pre-existing condition) that:

- 1. Was not present prior to the study, but appeared or reappeared following initiation of the study.
- 2. Was present prior to the study but worsened during the study. This would include any condition resulting from concomitant illnesses, reactions to concomitant medications, or progression of disease states.

**Note**: Pregnancy must be documented as an adverse event and must be reported to the clinical monitor and to the Sponsor immediately upon learning of the event.

Serious Adverse Event (SAE) – An SAE is any adverse event that led to any of the following:

- Death
- Serious deterioration in the health of the subject that resulted in any of the following:
- Life-threatening illness or injury
- Permanent or persistent impairment of a body structure or a body function
- Hospitalization or prolongation of patient hospitalization
- Medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function.
- Chronic disease
- Fetal distress, fetal death or a congenital physical or mental impairment of birth defect.

Diagnoses and conditions that are considered Ocular Serious Adverse Events include, but not limited to:

- Microbial Keratitis (MK)
- Iritis (including cells in the anterior chamber)
- Permanent decrease in best spectacle corrected visual acuity equivalent to 2 acuity lines or greater
- Central Corneal Opacity
- Central Corneal Neovascularization
- Uveitis
- Endophthalmitis
- Hypopyon
- Hyphemia
- Penetration of Bowman's Membrane
- Persistent Epithelial Defect
- Limbal cell Damage leading to Conjunctivalization

**Significant Adverse Events** – are defined as events that are symptomatic and warrant discontinuation (temporary or permanent) of the contact lens wear

Diagnoses and conditions that are considered Ocular Significant Adverse Events include, but not limited to the following:

- Contact Lens Induced Peripheral Ulcer (CLPU)
- Significant Infiltrative Events (SIE)
- Superior Epithelial Arcuate Lesions (SEALs)
- Any Temporary Loss of > 2 Lines of BSCVA
- Other grade 3 or higher corneal findings, such as abrasions or edema
- Non-contact lens related corneal events e.g. Epidemic Keratoconjunctivitis (EKC)
- Asymptomatic Corneal Scar
- Any corneal event which necessitates temporary lens discontinuation > 2 weeks

**Non-Significant Adverse Events** – are defined as those events that are usually asymptomatic and usually do not warrant discontinuation of contact lens wear but may cause a reduction in wear time. However, the Investigator may choose to prescribe treatment as a precautionary measure.

Diagnoses and conditions that are considered Ocular Non-Significant Adverse Events include, but not limited to the following:

- Non-significant Infiltrative Event (NSIE)
- Contact Lens Papillary Conjunctivitis (CLPC)
- Superficial Punctate Keratitis (SPK)
- Conjunctivitis: Bacterial, Viral, Allergic
- Blepharitis
- Meibomianitis
- Contact Dermatitis

- Localized Allergic Reactions
- Any corneal event not explicitly defined as serious or significant adverse event, which necessitates temporary lens discontinuation < 2 weeks

**Adverse Device Effect (ADE)** – An ADE is an "adverse event related to the use of an investigational medical device."

NOTE 1: This definition includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device.

NOTE 2: This definition includes any event resulting from use error or from intentional misuse of the investigational medical device.<sup>1</sup>

**Unanticipated Adverse Device Effect (UADE)** – A UADE is any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, the test article, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan, Investigator's Brochure or protocol, or any other unanticipated serious problem associated with the test article that relates to the rights, safety and welfare of subjects.

## 13.2. Assessing Adverse Events

In conjunction with the medical monitor, the Investigator will evaluate adverse events to ensure the events are categorized correctly. Elements of categorization will include:

- Seriousness/Classifications (see definition in section 13.1).
- Causality or Relatedness i.e. the relationship between the test article, study treatment or study procedures and the adverse event (not related, unlikely related, possibly related, or related see definition in section 13.2.1).
- Adverse Event Severity Adverse event severity is used to assess the degree of intensity of the adverse event (mild, moderate, or severe see definition in section 13.2.2).
- Outcome not recovered or not resolved, recovering or resolving, recovered or resolved with sequelae, recovered or resolved, death related to adverse event, or unknown.
- Actions Taken none, temporarily discontinued, permanently discontinued, or other.

### 13.2.1. Causality Assessment

Causality Assessment – A determination of the relationship between an adverse event and the test article. The test article relationship for each adverse event should be determined by the investigator using these explanations:

- Not Related- An adverse event that is not related to the use of the test article, study treatment or study procedures.
- Unlikely Related An adverse event for which an alternative explanation is more likely, e.g. concomitant treatment, concomitant disease(s), or the relationship of time suggests that a causal relationship is not likely.

- Possibly Related An adverse event that might be due to the use of the test article, or to the study treatment or study procedures. An alternative explanation, e.g. concomitant treatment, concomitant disease(s), is inconclusive. The relationship in time is reasonable. Therefore, the causal relationship cannot be excluded.
- Related An adverse event that is listed as a possible adverse effect (device) or adverse reaction (drug) and cannot be reasonably explained by an alternative explanation, e.g. concomitant treatment of concomitant disease(s). The relationship in time is very suggestive, e.g. it is confirmed by de-challenge and re-challenge.

### 13.2.2. Severity Assessment

**Severity Assessment** – A qualitative assessment of the degree of intensity of an adverse event as determined by the Investigator or reported to him/her by the subject. The assessment of severity is made irrespective of test article, study treatment or study procedure relationship or seriousness of the event and should be evaluated according to the following scale:

- Mild Event is noticeable to the subject but is easily tolerated and does not interfere with the subject's daily activities.
- Moderate Event is bothersome, possible requiring additional therapy, and may interfere with the subject's daily activities.
- Severe Event is intolerable, necessitates additional therapy or alteration of therapy and interferes with the subject's daily activities.

## 13.3. Documentation and Follow-Up of Adverse Events

The recording and documenting of adverse events (ocular and non-ocular) begin when the subjects are exposed to the test article, study treatment or study procedure. Adverse events reported before the use of test article, start of study treatment, or study procedures will be recorded as medical history. However, if the condition deteriorates at any time during the study, it will be recorded and reported as an AE. Untoward medical events reported after the subject's exit from the study will be recorded as adverse events at the discretion of the Investigator.

Upon finding an adverse event, the Principal Investigator will document the condition in the subject record and in the eCRFs and complete the Adverse Event eCRF.

Complete descriptions of all adverse events must be available in the subject record. All Adverse Events including local and systemic reactions not meeting the criteria for "serious adverse events" shall be captured on the appropriate case report form or electronic data system. All adverse events occurring while the subject is enrolled in the study must be documented appropriately regardless of relationship.

It is the Investigator's responsibility to maintain documentation of each reported adverse event. All adverse events will be followed in accordance with applicable licensing requirements. Such documentation will include the following:

- Adverse event (diagnosis not symptom).
- Drawings or photographs (where appropriate) that detail the finding (e.g., size, location, and depth, etc.).

- Date the clinical site was notified.
- Date and time of onset.
- Date and time of resolution.
- Adverse event classification, severity, and relationship to test articles, as applicable.
- Treatment regimen instituted (where appropriate), including concomitant medications prescribed, in accordance with applicable licensing requirements.
- Any referral to another health care provider if needed.
- Outcome, ocular damage (if any).
- Likely etiology.
- Best corrected visual acuity at the discovery of the event and upon conclusion of the event if the AE is related to the visual system.

Upon discovery of an AE that is deemed 'possibly related' or 'related' to the test article or study procedures (whether related to the visual system or not), an AE review form must be completed. Additional dated and initialed entries should be made at follow-up evaluations. Separate forms must be completed for each eye if the AE is bilateral.

In addition, if an infiltrate(s) is present, he/she will complete the Corneal Infiltrate Assessment eCRF. Where necessary, a culture of the corneal lesion will be collected to determine if the infection is microbial in nature. If cultures are collected, the date of culture collection and laboratory utilized will be recorded.

Changes in the severity of an AE shall be documented to allow an assessment of the duration of the event at each level of intensity to be performed. Adverse events characterized as intermittent require documentation of the onset and duration of each episode. Changes in the assessment of relationship to the Test Article shall also be clearly documented.

Subjects who present with an adverse event shall be followed by the Investigator, within licensure, until all signs and symptoms have returned to pre-treatment status, stabilized, or been satisfactorily resolved. If further treatment beyond licensure is required, the patient will be referred to the appropriate health care provider. The Investigator will use his/her clinical judgment as to whether a subject reporting with an adverse event will continue in the study. If a subject is discontinued from the study, it will be the responsibility of the Investigator to record the reason for discontinuation. The Investigator will also document the adverse event appropriately and complete the Adverse Event eCRF. Any subjects with ongoing adverse events related to the test article, study treatment or study procedures, as of the final study visit date, should be followed to resolution of the adverse event or until referral to an appropriate health care provider, as recommended by the Investigator. Non-ocular adverse events that are not related to the test article, study treatment, or study procedures may be recorded as "ongoing" without further follow-up.

### 13.4. Reporting Adverse Events

The Investigator will notify the Sponsor of an adverse event by e-mail, facsimile, or telephone as soon as possible and no later than 24 hours from discovery for any serious /significant adverse events, and 2 days from discovery for any non-significant adverse event. In addition,

a written report will be submitted by the Principal Investigator to the IEC/IRB according to their requirements (section 13.4.2). The report will comment whether the adverse event was considered to be related to the test article, study treatment or study procedures.

## 13.4.1. Reporting Adverse Events to Sponsor

## **Serious/Significant Adverse Events**

The Investigator will inform the sponsor of all serious/significant adverse events occurring during the study period as soon as possible by e-mail or telephone, but no later than 24 hours following discovery of the event. The Investigator is obligated to pursue and obtain information requested by the Sponsor in addition to that information reported on the eCRF. All subjects experiencing a serious/significant adverse event must be followed up and all outcomes must be reported.

When medically necessary, the Investigator may break the randomization code to determine the identity of the treatment that the subject received. The Sponsor and study monitor should be notified prior to unmasking the test articles.

In the event of a serious/significant adverse event, the Investigator must:

- Notify the Sponsor immediately.
- Obtain and maintain in the subject's records all pertinent medical information and medical judgment for colleagues who assisted in the treatment and follow-up of the subject.
- Provide the Sponsor with a complete case history which includes a statement as to whether the event was or was not related to the use of the test article.
- Notify the IEC/IRB as required by the IEC/IRB reporting procedure according to national regulations.

#### **Unanticipated (Serious) Adverse Device Effect (UADE)**

In the event of an Unanticipated (Serious) Adverse Device Effect (UADE), the Investigator will submit a report of the UADE to the Sponsor and IEC/IRB as soon as possible, but no later than 24 hours after the Investigator first learns of the effect. This report is in addition to the immediate notification mentioned above.

The Sponsor must conduct an evaluation of the UADE and must report the results of the evaluation to FDA, the IEC/IRB and participating Investigators within 10 working days after the Sponsor first receives notification of the effect.

#### **Non-Serious Adverse Events**

All non-serious adverse events, including non-serious adverse device effects, will be reported to the sponsor by the Investigator no later than 2 days from discovery.

### 13.4.2. Reporting Adverse Events to the Responsible IEC/IRB and Health Authorities

Adverse events that meet the IEC/IRB requirements for reporting must be reported within the IEC/IRB's written guidelines. Each clinical site will refer to and follow any guidelines set forth

by their Approving IEC/IRB. Each clinical site will refer to and follow any guidelines set forth by their local governing Health Authorities.

The Sponsor will report applicable Adverse Events to the local health authorities according to the written guidelines, including reporting timelines.

## 13.5. Event of Special Interest

None.

## 13.6. Reporting of Pregnancy

Subjects reporting pregnancy (by self-report) during the study will be discontinued after the event is recorded as an Adverse Event. Once discontinued, pregnant participants and their fetuses will not be monitored for study related purposes. Pregnant participants are not discontinued from contact lens or solution related studies for safety concerns, but due to general concerns relating to pregnancy and contact lens use. Specifically, pregnant women are discontinued due to fluctuations in refractive error and/or visual acuity that occur secondary to systemic hormonal changes, and not due to unforeseen health risks to the mother or fetus.

### 14. STATISTICAL METHODS

### 14.1. General Considerations

Statistical Analysis will be undertaken by the sponsor or under the authority of the sponsor. A general description of the statistical methods to be implemented in this clinical trial is outlined below.

All data summaries and statistical analyses will be performed using Statistical Analysis System (SAS) software Version 9.4 or higher (SAS Institute, Cary, NC). Throughout the analysis of data, the results for each subject/eye will be used when available for summarization and statistical analysis. Unscheduled visits will / will not be summarized separately and will / will not be excluded from the statistical analysis.

Summary tables (descriptive statistics and/or frequency tables) will be provided for all baseline variables, efficacy variables and safety variables as appropriate. Continuous variables will be summarized with descriptive statistics (n, mean, standard deviation (SD), median, minimum and maximum). Frequency count and percentage of subjects or eyes within each category will be provided for categorical data.

### 14.2. Sample Size Justification

The plan is to enroll 140 subjects with a target of at least 126 subjects to complete. The power calculation is based on 2-sequence and 3-period (Test/Control/Control or Control/Test/Test) crossover study design and study results from where prototype toric lens designs with the RTY-1 chromophore evaluated in a daily disposable modality against AO1DfA as control to demonstrate non-inferiority of the Test relative to the Control.

Table 6 provides a summary of power based on the primary hypothesis of non-inferiority for CLUE Comfort with 126 subjects to complete the study and two-sided Type I error of 0.05 with the assumptions for treatment effect (Test minus Control), standard deviation and intraclass correlation. The power calculation is conducted using 1000 simulations with linear mixed models using the GLIMMIX procedure in SAS 9.4.

Table 6: Power Calculation for the Primary Hypothesis of CLUE Comfort score (Non-inferiority of the Test relative to the Control) with Type I error of 0.05.

| Mean | | Number of Subjects (n/2 per sequence) | Within Subject Correlation | |
|---|---|---|---|---|
| Difference<br>(Test-Control) | Standard<br>Deviation | | 0.4 | 0.5 |
| -0.8 | 23 | 126 | 0.710 | 0.727 |
| -0.8 | 25 | 126 | 0.618 | 0.633 |
| 0 | 23 | 126 | 0.870 | 0.887 |
| 0 | 25 | 126 | 0.804 | 0.814 |
| 0.8 | 23 | 126 | 0.965 | 0.974 |
| 0.8 | 25 | 126 | 0.909 | 0.931 |

As shown in the Table 6, the study will be powered (power of 0.8 or higher) to show non-inferiority of the Test relative to the Control lens with respect to CLUE Comfort score when the mean difference  $\geq 0$ , the standard deviation  $\leq 25$  and an intraclass correlation  $\geq 0.4$ .

### 14.3. Analysis Populations

### Safety Population:

All subjects who are administered any test article excluding subjects who drop out prior to administering any test article. At least one observation should be recorded.

# Per-Protocol Population:

All subjects who successfully complete all visits and do not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock. Justification for the exclusion of subjects with protocol deviations from the Per-Protocol Population set will be documented in a memo to file.

## Intent-to-Treat (ITT) Population:

All randomized subjects regardless of actual treatment and subsequent withdrawal from the study or deviation from the protocol. At least one observation should be recorded.

# 14.4. Level of Statistical Significance

The primary analysis for this study will be conducted with an overall type I error rate of 5%. If any post-hoc statistical analysis after reviewing data is conducted, a type I error rate of 5% will be used for exploratory purposes.

# 14.5. Primary Analysis

#### **CLUE** Comfort score

CLUE Comfort scores at 1-week follow-up will be analyzed using a linear mixed effect model to compare between the Test and Control lenses. The model will include the baseline score, sequence, lens type, lens wearing period, and first order carryover effect as fixed effects. Additional fixed effects will include subject characteristics such as age and gender. Investigational site will be included as a random intercept. The covariance of residual errors between different periods for the same subject will be modeled using either homogenous compound symmetry (CS), heterogeneous compound-symmetry (HCS) or unstructured (UN) covariance structure. The structure that returns the lowest finite sample corrected Akaike's Information criterion will be selected as the structure that best fits the model. The Kenward and Roger method will be used for the calculation of the denominator degree of freedom.

The null and alternative hypotheses for non-inferiority of the Test - Control is as follows:

 $H_0$ :  $\Delta < -5$  $H_A$ :  $\Delta \ge -5$ 

where  $\Delta$  is the least square mean (LSM) difference of CLUE Comfort score at 1-week follow-up between the Test and Control lens (Test minus Control). Non-inferiority will be declared if the corresponding lower bound of the 95% two-sided confidence interval (CI) of the least squares mean (LSM) difference (Test - Control) for CLUE Comfort score at 1-week follow-up based on the per-protocol population is greater than -5.

### 14.6. Secondary Analysis

Not applicable.

## 14.7. Other Exploratory Analysis

Descriptive summary of the following efficacy endpoints by treatment arm will be provided on the per-protocol population.

- HLHC distance VA at the follow-up visit
- Settled lens orientation at the dispensing visit and at follow-up visits
- Lens rotational stability with blinks at the dispensing visit
- Subjective response to MRD questionnaire items at the follow-up visit
- Subjective response to the CLUE questionnaire Comfort, Vision, and Handling items at fitting

 Subjective response to the CLUE questionnaire Vision and Handling items at followup

# 14.8. Interim Analysis

Not applicable.

### 14.9. Procedure for Handling Missing Data and Drop-Outs

Missing or spurious values will not be imputed. The count of missing values will be included in the summary tables and listings.

### 14.10. Procedure for Reporting Deviations from Statistical Plan

The analysis will be conducted according to that specified in above sections. There are no known reasons for which it is planned to deviate from these analysis methods. If for any reason a change is made, the change will be documented in the study report along with a justification for the change.

#### 15. DATA HANDLING AND RECORD KEEPING/ARCHIVING

## 15.1. Electronic Case Report Form/Data Collection

The data for this study will be captured on electronic case report forms (eCRFs) using the BioClinica EDC system. An authorized data originator will enter study data into the eCRFs using the EDC system. Data collected on equipment that is not captured in EDC will be formatted to the specification of the JJVC database manager and sent to JJVC for analysis.

No external data sources will be included in this study.

The clinical data will be recorded on dedicated eCRFs specifically designed to match the study procedures for each visit. Only specifically delegated staff can enter data on a CRF. Once completed, the eCRFs will be reviewed for accuracy and completeness and signed by the Investigator. The sponsor or sponsor's representatives will be authorized to gain access to the subject recordation for the purposes of monitoring and auditing the study.

Edit checks, electronic queries, and audit trails are built into the system to ensure accurate and complete data collection. Data will be transmitted from the clinical site to a secure central database as forms are completed or updated, ensuring information accuracy, security, and confidentiality. After the final database lock, the Investigator will be provided with Individual Patient Profiles (IPP) including the full audit trail on electronic media in PDF format for all of the study data. The IPP must be retained in the study files as a certified copy of the source data for the study.

The content and structure of the eCRFs are compliant with ISO14155:2020.<sup>1</sup>

# 15.2. Subject Record

At a minimum, subject record should be available for the following:

- subject identification
- eligibility
- study identification
- study discussion
- provision of and date of informed consent
- visit dates
- results of safety and efficacy parameters as required by the protocol
- a record of all adverse events
- follow-up of adverse events
- medical history and concomitant medication
- test article receipt/dispensing/return records
- date of study completion
- reason for early discontinuation of test article or withdrawal from the study, if applicable

The subject record is the eCRF or an external record. The author of an entry in the subject record must be identifiable. The first point of entry is considered to be the source record.

Adverse event notes must be reviewed and initialed by the Investigator.

### 15.3. Trial Registration on ClinicalTrials.gov

This study will be registered on ClinicalTrials.gov by the Sponsor.

### 16. DATA MANAGEMENT

#### 16.1. Access to Source Data/Document

The Investigator/Institution will permit trial-related monitoring, audits, IEC/IRB review and regulatory inspection(s) by providing direct access to source data/documents. Should the clinical site be contacted for an audit by an IEC/IRB or regulatory authority, JJVC must be contacted and notified in writing within 24 hours.

# 16.2. Confidentiality of Information

Information concerning the investigational product and patent application processes, scientific data or other pertinent information is confidential and remains the property of JJVC. The Investigator may use this information for the purposes of the study only. It is understood by the Investigator that JJVC will use information developed in this clinical study in connection with the development of the investigational product and therefore may disclose it as required to other clinical investigators and to regulatory agencies. In order to allow the use of the information derived from this clinical study, the Investigator understands that he/she has an

obligation to provide complete test results and all data developed during this study to the Sponsor.

# 16.3. Data Quality Assurance

Steps will be taken to ensure the accuracy and reliability of data, include the selection of qualified investigators and appropriate clinical sites and review of protocol procedures with the Principal Investigator. The Principal Investigator, in turn, must ensure that all Sub-Investigators and clinical site personnel are familiar with the protocol and all study-specific procedures and have appropriate knowledge of the study article.

Training on case report form completion will be provided to clinical site personnel before the start of the study. The Sponsor will review case report forms for accuracy and completeness remotely during the conduct of the study, during monitoring visits, and after transmission to data management. Any data discrepancies will be resolved with the Investigator or designee, as appropriate.

Quality Assurance representatives from JJVC may visit clinical sites to review data produced during the study and to access compliance with applicable regulations pertaining to the conduct of clinical trials. The clinical sites will provide direct access to study-related source data/documents and reports for the purpose of monitoring and auditing by JJVC and for inspection by local and regulatory authorities.

# 16.4. Data Monitoring Committee (DMC)

Not applicable for this study.

#### 17. CLINICAL MONITORING

The study monitors will maintain close contact with the Principal Investigator and the Investigator's designated clinical site personnel. The monitor's responsibilities will include:

- Ensuring that the investigation is being conducted according to the protocol, any subsequent versions, and regulatory requirements are maintained.
- Ensuring the rights and wellbeing of subjects are protected.
- Ensuring adequate resources, including facilities, laboratories, equipment, and qualified clinical site personnel.
- Ensuring that protocol deviations are documented with corrective action plans, as applicable.
- Ensuring that the clinical site has sufficient test article and supplies.
- Clarifying questions regarding the study.
- Resolving study issues or problems that may arise.
- Reviewing of study records and source documentation verification in accordance with the monitoring plan.

#### 18. ETHICAL AND REGULATORY ASPECTS

# 18.1. Study-Specific Design Considerations

Potential subjects will be fully informed of the risks and requirements of the study and, during the study, subjects will be given any new information that may affect their decision to continue participation. Subjects will be told that their consent to participate in the study is voluntary and may be withdrawn at any time with no reason given and without penalty or loss of benefits to which they would otherwise be entitled. Subjects will only be enrolled if the fully able to understand the risks, benefits, and potential adverse events of the study and provide their consent voluntarily.

# 18.2. Investigator Responsibility

The Principal Investigator is responsible for ensuring that the clinical study is performed in accordance with the signed agreement, the investigational plan, section 4 of the ICH E6(R2) guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements. GCP is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human subjects. Compliance with this standard provides public assurance that the rights, safety, and well-being of study subjects are protected, consistent with the principles of the Declaration of Helsinki 64<sup>th</sup> WMA General Assembly 2013<sup>3</sup> and that the clinical study data are credible. The Investigator must maintain clinical study files in accordance with section 8 of the ICH E6(R2) guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements.

## 18.3. Independent Ethics Committee or Institutional Review Board (IEC/IRB)

Before the start of the study, the Investigator (or Sponsor when applicable) will provide the IEC/IRB with current and complete copies of the following documents (where applicable):

- Final protocol.
- Sponsor-approved informed consent form (and any other written materials to be provided to the subjects)
- Investigator's Brochure (or equivalent information).
- Sponsor-approved subject recruitment materials.
- Information on compensation for study-related injuries or payment to subjects for participation in the study.
- Investigator's curriculum vitae, clinical licenses, or equivalent information (unless not required, as documented by IEC/IRB).
- Information regarding funding, name of the Sponsor, institutional affiliations, other potential conflicts of interest, and incentives for subjects.
- Any other documents that the IEC/IRB requests to fulfill its obligation.

This study will be undertaken only after IEC/IRB has given full approval of the final protocol, the informed consent form, applicable recruiting materials, and subject compensation programs, and the Sponsor has received a copy of this approval. This approval letter must be dated and must clearly identify the documents being approved.

During the study, the Investigator (or Sponsor when applicable) will send the following documents to the IEC/IRB for their review and approval, where appropriate:

- Protocol revisions
- Revision(s) to informed consent form and any other written materials to be provided to subjects
- If applicable, new or revised subject recruitment materials approved by the Sponsor
- Revisions to compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's Brochure revisions
- Summaries of the status of the study (at least annually or at intervals stipulated in guidelines of the IEC/IRB)
- Reports of adverse events that are serious, unanticipated, and associated with the test articles, according to the IRB's requirements
- New information that may adversely affect the safety of the subjects or the conduct of the study
- Major protocol deviations as required by the IEC/IRB
- Report of deaths of subjects under the Investigator's care
- Notification if a new Investigator is responsible for the study at the clinical site
- Any other requirements of the IEC/IRB

For protocol revisions that increase subject risk, the revisions and applicable informed consent form revisions must be submitted promptly to the IEC/IRB for review and approval before implementation of the change(s).

At least once a year, the IEC/IRB will review and reapprove this clinical study. This request should be documented in writing.

At the end of the study, the Investigator (or Sponsor where required) will notify the IEC/IRB about the study completion. Documentation of this notification must be retained at the clinical site and a copy provided to the CRO or Sponsor as applicable.

### 18.4. Informed Consent

Each subject or their representative, must give written consent according to local requirements after the nature of the study has been fully explained. The consent form must be signed before performance of any study-related activity. The consent form that is used must be approved by both the Sponsor and by the reviewing IEC/IRB. The informed consent is in accordance with principles that originated in the Declaration of Helsinki,<sup>3</sup> current ICH GCP<sup>2</sup> and ISO 14155:2020<sup>1</sup> guidelines, applicable regulatory requirements, and Sponsor Policy.

Before entry into the study, the Investigator or an authorized member of the clinical site personnel must explain to potential subject the aims, methods, reasonably anticipated benefits, and potential hazards of the study, and any discomfort it may entail. Subjects will be informed that their participation is voluntary and that they may withdraw consent to participate at any time.

The subject will be given sufficient time to read the informed consent form and the opportunity to ask questions. After this explanation and before entry into the study, consent should be appropriately recorded by means of the subject's dated signature. After having obtained the consent, a copy of the informed consent form must be given to the subject.

### 18.5. Privacy of Personal Data

The collection, processing and disclosure of personal data and medical information related to the Study Subject, and personal data related to Principal Investigator and any clinical site personnel (e.g., name, clinic address and phone number, curriculum vitae) is subject to compliance with the Health Information Portability and Accountability Act (HIPAA) in the United States<sup>7</sup> and other applicable personal data protection and security laws and regulations. Appropriate measures will be employed to safeguard these data, to maintain the confidentiality of the person's related health and medical information, to properly inform the concerned persons about the collection and processing of their personal data, to grant them reasonable access to their personal data and to prevent access by unauthorized persons.

All information obtained during the course of the investigation will be regarded as confidential. All personal data gathered in this trial will be treated in strictest confidence by Investigators, monitors, Sponsor's personnel and IEC/IRB. No data will be disclosed to any third party without the express permission of the subject concerned, with the exception of Sponsor personnel (monitor, auditor), IEC/IRB and regulatory organizations in the context of their investigation related activities that, as part of the investigation will have access to the CRFs and subject records.

The collection and processing of personal data from subjects enrolled in this study will be limited to those data that are necessary to investigate the efficacy, safety, quality, and utility of the investigational product(s) used in this study.

These data must be collected and processed with adequate precautions to ensure confidentiality and compliance with applicable data privacy protection laws and regulations.

The Sponsor ensures that the personal data will be:

- processed fairly and lawfully.
- collected for specified, explicit, and legitimate purposes and not further processed in a way incompatible with these purposes.
- adequate, relevant, and not excessive in relation to said purposes.
- accurate and, where necessary, kept current.

Explicit consent for the processing of personal data will be obtained from the participating subject before collection of data. Such consent should also address the transfer of the data to other entities and to other countries.

The subject has the right to request through the Investigator access to his personal data and the right to request rectification of any data that are not correct or complete. Reasonable steps should be taken to respond to such a request, taking into consideration the nature of the request, the conditions of the study, and the applicable laws and regulations.

Appropriate technical and organizational measures to protect the personal data against unauthorized disclosures or access, accidental or unlawful destruction, or accidental loss or alteration must be put in place. Sponsor personnel whose responsibilities require access to personal data agree to keep the identity of study subjects confidential.

### 19. STUDY RECORD RETENTION

In compliance with the ICH GCP guidelines,<sup>2</sup> the Investigator/Institution will maintain all CRFs and all subject records that support the data collected from each subject, as well as all study documents as specified in ICH GCP<sup>2</sup> and all study documents as specified by the applicable regulatory requirement(s). The Investigator/Institution will take measures to prevent accidental or premature destruction of these documents.

Essential documents must be retained until at least two (2) years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or until at least two (2) years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period if required by the applicable regulatory requirements or instructed by the Sponsor. It is the responsibility of the Sponsor to inform the Investigator/Institution as to when these documents no longer need to be retained.

If the responsible Investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will accept the responsibility. The Sponsor must be notified in writing of the name and address of the new custodian. Under no circumstance shall the Investigator relocate or dispose of any study documents before having obtained written approval from the Sponsor.

If it becomes necessary for the Sponsor or the appropriate regulatory authority to review any documentation relating to this study, the Investigator must permit access to such reports. If the Investigator has a question regarding retention of study records, he/she should contact JJVC.

### 20. FINANCIAL CONSIDERATIONS

Remuneration for study services and expenses will be set forth in detail in the Clinical Research Agreement. The Research Agreement will be signed by the Principal Investigator and a JJVC management representative prior to study initiation.

JJVC reserves the right to withhold remuneration for costs associated with protocol violations such as:

- Continuing an ineligible subject in the study.
- Scheduling a study visit outside the subject's acceptable visit range.

JJVC reserves the right to withhold final remuneration until all study related activities have been completed, such as:

- Query resolution.
- Case Report Form signature.
- Completion of any follow-up action items.

### 21. PUBLICATION

There is no plan to externally publish this outcome of this investigation.

#### 22. REFERENCES

- 1. ISO 14155:2020: Clinical Investigation of Medical Devices for Human Subjects Good Clinical Practice. Available at: https://www.iso.org/standard/71690.html
- 2. International Council for Harmonization Good Clinical Practice E6(R2) (ICH GCP). Available at: https://www.ich.org/page/efficacy-guidelines
- 3. Declaration of Helsinki Ethical principles for Medical Research Involving Human Subjects. Available at: https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects/
- 4. United States (US) Code of Federal Regulations (CFR). Available at: https://www.gpo.gov/fdsys/browse/collectionCfr.action?collectionCode=CFR
- 5. Straker B. Investigator's Brochure: Toric lens design in senofilcon A with HEV-blocking chromophore (RTY-1). 2022.
- 6. Wirth RJ, et al. Development of the contact lens user experience: CLUE scales. *Optometry and Vision Science*. 2016;93.8:801.
- 7. Health Information Portability and Accountability Act (HIPAA). Available at: https://www.hhs.gov/hipaa/for-professionals/privacy/index.html
- 8. Keselman HJ, Algina J, Kowalchuk RK, Wolfinger RD. A comparison of two approaches for selecting covariance structures in the analysis of repeated measurements. *Communications in Statistics Simulation and Computation*. 1998;27(3):591-604.
- 9. Kenward MG, Roger JH. Small Sample Inference for Fixed Effects from Restricted Maximum Likelihood. *Biometrics*. 1997;53(3):983.

APPENDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES)











# Clinical Study Protocol Johnson & Johnson Vision Care, Inc.

#### APPENDIX B: PATIENT INSTRUCTION GUIDE

Will be provided separately.

# Clinical Study Protocol Johnson & Johnson Vision Care, Inc.

APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT)

ACUVUE Oasys 1-Day for Astigmatism

IMPORTANT: Please read carefully and keep this information for future use.

This Package Insert and Fitting Guide is intended for the Eye Care Professional, but should be made available to patients upon request.

The Eye Care Professional should provide the patient with the appropriate instructions that pertain to the patient's prescribed lenses. Copies are available for download at www.acuvue.com.



ACUVUE OASYS® Brand Contact Lenses 1-Day with HydraLuxe™ Technology

ACUVUE OASYS® Brand Contact Lenses 1-Day with HydraLuxe™ Technology for ASTIGMATISM

senofilcon A Soft (hydrophilic) Contact Lenses Visibility Tinted with UV Blocker for Daily Disposable Wear




# SYMBOLS KEY

The following symbols may appear on the label or carton:

| SYMBOL | DEFINITION |
|---|---|
| i | Consult Instructions for Use |
| | Manufactured by or in |
| | Date of Manufacture |
| $\subseteq$ | Use By Date (expiration date) |
| LOT | Batch Code |
| STERILE | Sterile Using Steam or Dry Heat |
| 2 | Single-Use |
| DIA | Diameter |
| ВС | Base Curve |
| D | Diopter (lens power) |
| CYL | Cylinder |
| AXIS | Axis |
| <b>C€</b><br>0086 | Quality System Certification Symbol |
| UV Blocking | UV-Blocking |
| • | Fee Paid for Waste Management |
| <b>R</b> Only | CAUTION: U.S. Federal law restricts this device to sale by or on the order of a licensed practitioner |
| 123 💙 | Lens Orientation Correct |
| X X | Lens Orientation Incorrect (Lens Inside Out) |

CR-6484, v 1.0

#### **DESCRIPTION**

ACUVUE OASYS® Brand Contact Lenses 1-Day and ACUVUE OASYS® Brand Contact Lenses 1-Day for ASTIGMATISM are soft (hydrophilic) contact lenses made with HydraLuxe<sup>TM</sup> Technology. They are available as spherical or toric lenses respectively.

These lenses are made of a silicone hydrogel material containing an internal wetting agent, visibility tint, and UV absorbing monomer and are tinted blue using Reactive Blue Dye #4 to make the lenses more visible for handling.

A benzotriazole UV absorbing monomer is used to block UV radiation. The transmittance characteristics for these lenses are less than 1% in the UVB range of 280 nm to 315 nm and less than 10% in the UVA range of 316 nm to 380 nm for the entire power range.

#### Lens Properties:

#### The physical/optical properties of the lens are:

| <ul> <li>Specific Gravity (calculated):</li> </ul> | 0.98 - | 1.12 |
|----------------------------------------------------|--------|------|
|----------------------------------------------------|--------|------|

Refractive Index: 1.42

Light Transmission:
 85% minimum

Surface Character: Hydrophilic

• Water Content: 38%

Oxygen Permeability:

| <b>VAL</b> | _UE | METHOD |
|------------|-----|--------|

 $122 \times 10^{-11} \text{ (cm}^2\text{/sec)} \qquad \qquad \text{Fatt (boundary corrected, non-model} \\ \text{(ml O}_2/\text{ml x mm Hg) at } 35^{\circ}\text{C} \qquad \qquad \text{edge corrected)} \\ 103 \times 10^{-11} \text{ (cm}^2\text{/sec)} \qquad \qquad \text{Fatt (boundary corrected, edge (ml O}_2/\text{ml x mm Hg) at } 35^{\circ}\text{C} \qquad \qquad \text{corrected)} \\ \end{cases}$ 

#### **Lens Parameters:**

Diameter Range: 12.0 mm to 15.0 mm
Center Thickness: varies with power
Base Curve Range: 7.85 mm to 10.00 mm
Spherical Power Range: -20.00D to +20.00D

• Cylinder Power Range: -0.25D to -10.00D

Axis Range: 5° to 180° CONFIDENTIAL


#### **AVAILABLE LENS PARAMETERS**

ACUVUE OASYS® Brand 1-Day with HydraLuxe™ Technology are hemispherical shells of the following dimensions:

**Diameter:** 14.3 mm

**Center Thickness:** 0.085 mm to 0.221 mm (varies with power)

**Base Curve:** 8.5 mm. 9.0 mm

**Powers:** -0.50D to -6.00D (in 0.25D increments)

-6.50D to -12.00D (in 0.50D increments) +0.50D to +6.00D (in 0.25D increments) +6.50D to +8.00D (in 0.50D increments)

ACUVUE OASYS® Brand 1-Day with HydraLuxe™ Technology for ASTIGMATISM are hemitoric shells of the following dimensions:

**Diameter:** 14.3 mm

**Center Thickness:** 0.075 mm to 0.172 mm (varies with power)

**Base Curve:** 8.5 mm

**Powers:** +0.00D to -6.00D (in 0.25D increments)

Cylinders: -0.75D, -1.25D, -1.75D, -2.25D\*

Axis: 10° to 180° in 10° increments

\*-2.25D cylinder is available in 10°, 20°, 70°, 80°, 90°, 100°, 110°,

160°, 170°, 180° axes only.

+0.25D to +4.00D (in 0.25D increments)

-6.50D to -9.00D (in 0.50D increments)

Cylinders: -0.75D, -1.25D, -1.75D

Axis: 10°, 20°, 70°, 80°, 90°, 100°, 110°, 160°,

170°, 180°

# TRANSMITTANCE CURVES

ACUVUE OASYS® 1-Day with HydraLuxe™ Technology (senofilcon A) Visibility Tinted with UV Blocker vs. 24 yr. old human cornea and 25 yr. old human crystalline lens.



<sup>\*</sup> The data was obtained from measurements taken through the central 3-5 mm portion for the thinnest marketed lens (-9.00D lens, 0.075 mm center thickness).

<sup>1</sup>Lerman, S., Radiant Energy and the Eye, MacMillan, New York, 1980, p. 58, figure 2-21

<sup>2</sup>Waxler, M., Hitchins, V.M., Optical Radiation and Visual Health, CRC Press, Boca Raton, Florida, 1986, p. 19, figure 5

WARNING: UV absorbing contact lenses are NOT substitutes for protective UV absorbing eyewear, such as UV absorbing goggles or sunglasses because they do not completely cover the eye and surrounding area. The patient should continue to use UV absorbing eyewear as directed.

#### **ACTIONS**

In its hydrated state, the contact lens, when placed on the cornea, acts as a refracting medium to focus light rays onto the retina.

The transmittance characteristics for these lenses are less than 1% in the UVB range of 280 nm to 315 nm and less than 10% in the UVA range of 316 nm to 380 nm for the entire

NOTE: Long-term exposure to UV radiation is one of the risk factors associated with cataracts. Exposure is based on a number of factors such as environmental conditions (altitude, geography, cloud cover) and personal factors (extent and nature of outdoor activities). UV-Blocking contact lenses help provide protection against harmful UV radiation. However, clinical studies have not been done to demonstrate that wearing UV-Blocking contact lenses reduces the risk of developing cataracts or other eye disorders. The Eye Care Professional should be consulted for more information.

# **INDICATIONS (USES)**

ACUVUE OASYS® Brand Contact Lenses 1-Day with HydraLuxe™ Technology are indicated for daily disposable wear for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes who may have 1.00D or less of astigmatism.

ACUVUE OASYS® Brand Contact Lenses 1-Day with HydraLuxe™ Technology for ASTIGMATISM are indicated for daily disposable wear for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes who may have 0.50D to 3.00D of astigmatism.

These lenses contain a UV Blocker to help protect against transmission of harmful UV radiation to the cornea and into the eye.

# **CONTRAINDICATIONS (REASONS NOT TO USE)**

# DO NOT USE these contact lenses when any of the following conditions exist:

- Acute or subacute inflammation or infection of the anterior chamber of the eye.
- Any eye disease, injury or abnormality that affects the cornea, conjunctiva, or eyelids.
- Severe insufficiency of lacrimal secretion (dry eye).
   CR-6484, v 1.0
   JJVC CONFIDENTIAL

- Corneal hypoesthesia (reduced corneal sensitivity).
- Any systemic disease that may affect the eye or be exaggerated by wearing contact lenses.
- Allergic reactions of ocular surfaces or adnexa that may be induced or exaggerated by wearing contact lenses or use of contact lens solutions.
- Ocular irritation due to allergic reactions which may be caused by use of contact lens solutions (i.e., rewetting drops) that contain chemicals or preservatives (such as mercury, Thimerosal, etc.) to which some people may develop an allergic response.
- Any active corneal infection (bacterial, fungal, protozoal, or viral).
- If eyes become red or irritated.

#### **WARNINGS**

Patients should be advised of the following warnings pertaining to contact lens wear:

EYE PROBLEMS, INCLUDING CORNEAL ULCERS, CAN DEVELOP RAPIDLY AND LEAD TO LOSS OF VISION; IF THE PATIENT EXPERIENCES:

- Eye Discomfort,
- Excessive Tearing,
- Vision Changes,
- Loss of Vision,
- Eye Redness,
- Or Other Eye Problems,

THE PATIENT SHOULD BE INSTRUCTED TO IMMEDIATELY REMOVE THE LENSES AND PROMPTLY CONTACT THE EYE CARE PROFESSIONAL.

When prescribed for daily wear, patients should be instructed not to wear lenses while sleeping. Clinical studies have shown that the risk of serious advers actions is increased when lenses are worn overnight, and that


extended wear contact lens users than for daily wear users.3

- Studies have shown that contact lens wearers who are smokers have a higher incidence of adverse reactions than nonsmokers.
- Problems with contact lenses or lens care products could result in serious injury to the eye. Patients should be cautioned that proper use and care of contact lenses and lens care products are essential for the safe use of these products.
- The overall risk of ulcerative keratitis may be reduced by carefully following directions for lens care.

#### **Specific Instructions for Use and Warnings:**

Water Activity

#### **Instructions for Use**

Do not expose contact lenses to water while wearing them.

#### **WARNING:**

Water can harbor microorganisms that can lead to severe infection, vision loss or blindness. If lenses have been submersed in water when participating in water sports or swimming in pools, hot tubs, lakes, or oceans, the patient should be instructed to discard them and replace them with a new pair. The Eye Care Professional should be consulted for recommendations regarding wearing lenses during any activity involving water.

# **PRECAUTIONS**

## **Special Precautions for Eye Care Professionals:**

Due to the small number of patients enrolled in clinical investigation of lenses, all refractive powers, design configurations, or lens parameters available in the lens material are not evaluated in significant numbers. Consequently, when selecting an appropriate lens design and parameters, the Eye Care Professional should consider all characteristics of the lens that can affect lens performance and ocular health, including oxygen permeability, wettability, central and peripheral thickness, and optic zone diameter.

<sup>&</sup>lt;sup>3</sup> New England Journal of Medicine, September 21, 1989; 321 (12), pp. 773-783

- The potential impact of these factors on the patient's ocular health should be carefully weighed against the patient's need for refractive correction; therefore, the continuing ocular health of the patient and lens performance on the eye should be carefully monitored by the prescribing Eye Care Professional.
- Patients who wear these lenses to correct presbyopia using monovision may not achieve the best corrected visual acuity for either far or near vision. Visual requirements vary with the individual and should be considered when selecting the most appropriate type of lens for each patient.
- Fluorescein, a yellow dye, should not be used while the lenses are
  on the eyes. The lenses absorb this dye and become discolored.
  Whenever fluorescein is used in eyes, the eyes should be flushed
  with a sterile saline solution that is recommended for in-eye use.
- Eye Care Professionals should instruct the patient to remove the lenses immediately if the eyes become red or irritated.

# Eye Care Professionals should carefully instruct patients about the following care regimen and safety precautions.

#### **Handling Precautions:**

- Before leaving the Eye Care Professional's office, the patient should be able to promptly remove the lenses or should have someone else available who can remove the lenses for him or her.
- DO NOT use if the sterile blister package is opened or damaged.
- Always wash and rinse hands before handling lenses. Do not get cosmetics, lotions, soaps, creams, deodorants, or sprays in the eyes or on the lenses. It is best to put on lenses before putting on makeup. Water-based cosmetics are less likely to damage lenses than oil-based products.
- DO NOT touch contact lenses with the fingers or hands if the hands are not free of foreign materials, as microscopic scratches of the lenses may occur, causing distorted vision and/or injury to the eye.
- Carefully follow the handling in rt n, removal and wearing instructions in the "Patient of the Dage 88 of 170

wearing schedule and those prescribed by the Eye Care Professional.

- Always handle lenses carefully and avoid dropping them.
- Never use tweezers or other tools to remove lenses from the lens container unless specifically indicated for that use. Slide the lens up the side of the bowl until it is free of the container.
- Do not touch the lens with fingernails.

#### **Lens Wearing Precautions:**

- If the lens sticks (stops moving) on the eye, follow the recommended directions in "Care for a Sticking (Non-Moving) Lens." The lens should move freely on the eye for the continued health of the eye. If non-movement of the lens continues, the patient should be instructed to immediately consult his or her Eye Care Professional.
- Never wear lenses beyond the period recommended by the Eye Care Professional.
- The patient should be advised to never allow anyone else to wear their lenses. They have been prescribed to fit their eyes and to correct their vision to the degree necessary. Sharing lenses greatly increases the chance of eye infections.
- If aerosol products, such as hair spray, are used while wearing lenses, exercise caution and keep eyes closed until the spray has settled.
- Avoid all harmful or irritating vapors and fumes while wearing lenses.
- Always discard lenses worn as prescribed by the Eye Care Professional.

#### **Lens Care Precautions:**

 The patient should be informed that no cleaning or disinfection is needed when lenses are worn for daily disposable wear. Patients should always dispose of lenses when removed and have spare lenses or spectacles available.

#### Other Topics to Discuss with Patients:

- Always contact the Eye Care Professional before using any medicine in the eyes.
- Certain medications, such as antihistamines, decongestants, diuretics, muscle relaxants, tranquilizers, and those for motion sickness may cause dryness of the eye, increased lens awareness, or blurred vision. Should such conditions exist, proper remedial measures should be prescribed. Depending on the severity, this could include the use of lubricating drops that are indicated for use with soft contact lenses or the temporary discontinuance of contact lens wear while such medication is being used.
- Oral contraceptive users could develop visual changes or changes in lens tolerance when using contact lenses. Patients should be cautioned accordingly.
- As with any contact lens, follow-up visits are necessary to assure the continuing health of the patient's eyes. The patient should be instructed as to a recommended follow-up schedule.

#### Who Should Know That the Patient is Wearing Contact Lenses?

- Patients should inform all doctors (Health Care Professionals) about being a contact lens wearer.
- Patients should always inform their employer of being a contact lens wearer. Some jobs may require use of eye protection equipment or may require that the patient not wear contact lenses.

# **ADVERSE REACTIONS**

# The patient should be informed that the following problems may occur when wearing contact lenses:

- The eye may burn, sting, and/or itch.
- There may be less comfort than when the lens was first placed on the eye.
- There may be a feeling of something in the eye (foreign body, scratched area).
- There may be the potenti e temporary impairment due to

  
peripheral infiltrates, peripheral corneal ulcers, or corneal erosion. There may be the potential for other physiological observations, such as local or generalized edema, corneal neovascularization, corneal staining, injection, tarsal abnormalities, iritis, and conjunctivitis; some of which are clinically acceptable in low amounts.

- There may be excessive watering, unusual eye secretions, or redness of the eye.
- Poor visual acuity, blurred vision, rainbows, or halos around objects, photophobia, or dry eyes may also occur if the lenses are worn continuously or for too long a time.

The patient should be instructed to conduct a simple 3-part self-examination at least once a day. They should ask themselves:

- How do the lenses feel on my eyes?
- How do my eyes look?
- Have I noticed a change in my vision?

If the patient reports any problems, he or she should be instructed to IMMEDIATELY REMOVE THE LENS. If the problem or discomfort stops, the patient should discard the lens and place a new fresh lens on the eye.

If after inserting the new lens, the problem continues, the patient should be directed to IMMEDIATELY REMOVE THE LENS AND CONTACT HIS OR HER EYE CARE PROFESSIONAL.

The patient should be instructed NOT to use a new lens as self-treatment for the problem.

The patient should be advised that when any of the above symptoms occur, a serious condition such as infection, corneal ulcer, neovascularization, or iritis may be present. He or she should be instructed to seek immediate professional identification of the problem and prompt treatment to avoid serious eye damage.



#### **GENERAL FITTING GUIDELINES**

#### A. Patient Selection

Patients selected to wear these lenses should be chosen based on:

- Motivation to wear lenses
- Ability to follow instructions regarding lens wear care
- General health
- Ability to adequately handle and care for the lenses
- Ability to understand the risk and benefits of lens wear

Patients who do not meet the above criteria should not be provided with contact lenses.

#### B. Pre-fitting Examination

Initial evaluation of the patient should begin with a thorough case history to determine if there are any contraindications to contact lens wear. During the case history, the patient's visual needs and expectations should be determined as well as an assessment of their overall ocular, physical, and mental health.

Preceding the initial selection of trial contact lenses, a comprehensive ocular evaluation should be performed that includes, but is not limited to, the measurement of distance and near visual acuity, distance and near refractive prescription (including determining the preferred reading distance for presbyopes), keratometry, and biomicroscopic evaluation.

Based on this evaluation, if it is determined that the patient is eligible to wear these lenses, the Eye Care Professional should proceed to the lens fitting instructions as outlined below.

#### C. Initial Power Determination

A spectacle refraction should be performed to establish the patient's baseline refractive status and to guide in the selection of the appropriate lens power. Remember to compensate for vertex distance if the refraction is greater than  $\pm 4.00 \text{D}.$ 

#### D. Base Curve Selection (Trial Lens Fitting)

The following trial lenses should be selected for patients regardless of keratometry readings. However, the patient's baseline occlar status.


- ACUVUE OASYS® 1-Day: 8.5 mm/14.3 mm
- ACUVUE OASYS® 1-Day for ASTIGMATISM: 8.5 mm/14.3 mm

The trial lens should be placed on each of the patient's eyes and evaluated after the patient has adjusted to the lenses.

#### 1. Criteria of a Properly Fit Lens

A properly fit lens will center and completely cover the cornea (i.e., no limbal exposure), have sufficient movement to provide tear exchange under the contact lens with the blink, and be comfortable. The lens should move freely when manipulated digitally with the lower lid, and then return to its properly centered position when released.

#### 2. Criteria of a Flat Fitting Lens

A flat fitting lens may exhibit one or more of the following characteristics: decentration, incomplete corneal coverage (i.e., limbal exposure), excessive movement with the blink, and/or edge standoff. If the lens is judged to be flat fitting, it should not be dispensed to the patient.

#### 3. Criteria of a Steep Fitting Lens

A steep fitting lens may exhibit one or more of the following characteristics: insufficient movement with the blink, conjunctival indentation, and resistance when pushing the lens up digitally with the lower lid. If the lens is judged to be steep fitting, it should not be dispensed to the patient.

If the initial trial base curve is judged to be flat or steep fitting, the alternate base curve, if available, should be trial fit and evaluated after the patient has adjusted to the lens. The lens should move freely when manipulated digitally with the lower lid, and then return to a properly centered position when released. If resistance is encountered when pushing the lens up, the lens is fitting tightly and should not be dispensed to the patient.

#### E. Final Lens Power (Spherical)

A spherical over-refraction should be performed to determine the final lens power after the lens fit is judged acceptable. The spherical over-refraction should be combined with the trial lens power to determine the final lens prescription of the patient should prescription and prescription of the final lens power unless there are good, visual action at the correct lens power unless there are some of the final lens power unless there are some of the final lens power to determine the final lens prescription.


| Example 1 | |
|----------------------------|--------|
| Diagnostic lens: | -2.00D |
| Spherical over-refraction: | -0.25D |
| Final lens power: | -2.25D |

| Example 2 | |
|----------------------------|--------|
| Diagnostic lens: | -2.00D |
| Spherical over-refraction: | +0.25D |
| Final lens power: | -1.75D |

If vision is acceptable, perform a slit lamp examination to assess adequate fit (centration and movement). If the fit is acceptable, dispense the lenses and instruct the patient to return in one week for reassessment (see dispensing and follow up information in **PATIENT MANAGEMENT**).

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

#### TORIC FITTING GUIDELINES

Although most aspects of the fitting procedure are identical for all types of soft contact lenses, including toric lenses, there are some additional steps and/or rules to follow to assure the proper fit of toric lenses.

The only new steps you must follow in prescribing ACUVUE OASYS® 1-Day for ASTIGMATISM are that you must determine the stability, repeatability, and drift angle of the lens axis so that you can prescribe the correct lens axis for the patient.

#### A. How to Determine Lens Cylinder and Axis Orientation

#### 1. Locate the Orientation Marks

To help determine the proper orientation of the toric lens, you'll find two primary marks approximately 1 mm from the lens edge representing the vertical position on opposite ends of the lens at 6 and 12 o'clock (Fig. 1). Because of the lens' ballasting system, either mark can represent the vertical position – there is no "top" and "bottom" as in a prism-ballasted lens. You don't need to view both marks to assess orientation; simply look for the 6 o'clock mark as you would with a prism-ballasted lens.




You'll need a slit lamp biomicroscope with a 1 to 2 mm parallelepiped beam to highlight the marks when the lens is fitted to the eye. There are a number of techniques you can use to improve the visibility of the 6 o'clock mark. Using a parallelepiped beam and medium magnification (10x or 15x), slowly pan down the lens, looking just below the direct illumination at the retroilluminated area. Backlighting the mark this way should make it more visible. Sometimes manipulating the lower lid may be necessary to uncover the mark.

#### 2. Observe Lens Rotation and Stability

Observe the position and stability of the "bottom" mark. It usually stabilizes at the 6 o'clock position. If it does, calculation of the lens power will be straightforward. The 6 o'clock position is not a "must"; however, the absolute requirement is that the axis position be stable and repeatable.

The mark may stabilize somewhat left or right (drift) of the vertical meridian and still enable you to fit a toric lens for that eye, as long as the lens always returns to the same "drift axis" position after settling. The deviation can be compensated for in the final prescription. Your objective is to ensure that whatever position the initial lens assumes near 6 o'clock, this position must be stable and repeatable. With full eye movement or heavy blink, you may see the marks swing away, but they must return quickly to the original stable position. If the lens does not return quickly, you may need to select a different lens.

## 3. Assessing Rotation

Imagine the eye as a clock dial and every hour represents a 30° interval. If the orientation mark of the initial lens stabilizes somewhat left or right of the vertical position, the final lens will orient on the eye with the same deviation. You can use an axis reticule in the slit lamp or use a line-scribed lens in a spectacle trial frame to measure or estimate the "drift angle" of the cylinder axis.

To compensate for this "drift", measure or estimate the "drift", then add or subtract it from the refractive axis to determine the correct cylinder axis. Use the LARS (Left Add, Right Subtract) method to determine which direction to compensate.

#### **B. Final Lens Power**

When the diagnostic lens has its axis aligned in the same meridian as the patient's refractive axis, a spherocylindrical over-refraction may be performed and visual acuity determined. However, in the case of crossed axes, such as when the diagnostic lens axis is different from the spectacle cylinder axis, it is not advisable to perform a full spherocylindrical over-refraction because of the difficulty in computing the resultant power. A spherical over-refraction without cylinder refraction may be performed.

If the required cylinder correction falls between two available cylinder powers, it is recommended to prescribe the lower cylinder power lens. See below for instructions on how to determine the final lens power.

#### 1. For the Sphere

If sphere alone or combined sphere and cylinder Rx  $> \pm 4.00$ D, compensate for vertex distance. If sphere alone or combined sphere and cylinder Rx  $\leq \pm 4.00$ D, vertex compensation is not necessary.

#### 2. For the Cylinder

Adjust the axis by the drift angle using the LARS method. Choose a cylinder that is  $\leq$  0.50D from the refractive cylinder.

#### 3. Case Examples

## Example 1

Manifest (spectacle) refraction:

O.D. -2.50D / -1.25D x 180° 20/20

O.S. -2.00D / -1.00D x 180° 20/20

Choose a diagnostic lens for each eye with axis 180°. Place the lens on each eye and allow a minimum of 3 minutes for it to equilibrate, based on the patient's initial response to the lens. If the lens has not yet stabilized, recheck until stable.

Check the orientation of the axis mark. If the bottom axis mark is in the 6 o'clock position on both eyes, choose the appropriate cylinder as listed previously. If the lens has not yet stabilized, recheck until stable.

Here is the Rx Prescribed:

O.D. -2.50D / -1.25D x 180°

O.S. -2.00D / -0.75D x 180°

CR-6484, v 1.0



#### Example 2

Manifest (spectacle) refraction: O.D. -3.00D / -1.00D x 90° 20/20 O.S. -4.75D / -2.00D x 90° 20/20

Choose diagnostic lenses of -3.00D / -0.75D x 90° for the right eye and -4.50D / -1.75D x 90° for the left eye, the nearest lenses available to the spherical power, cylinder power, and axis needed. For the left eye, since the manifest refraction called for -4.75D, compensating for vertex distance the sphere is reduced by 0.25D to -4.50D. The cylinder power will be -1.75D. Place the lens on each eye and allow a minimum of 3 minutes for it to equilibrate, based on the patient's initial response to the lens. If the lens has not yet stabilized, recheck until stable.

#### Right Eye

The orientation mark on the right lens rotates left from the 6 o'clock position by 10° and remains stable in this position. Compensation for this rotation should be done as follows:

Compensate the 10° axis drift by adding it to the manifest refraction axis.

Here is the Rx Prescribed: O.D. -3.00D / -0.75D x 100°

#### Left Eye

The orientation mark on the left lens rotates right from the 6 o'clock position by 10° and remains stable in this position.

Compensate for the 10° axis drift by subtracting it from the manifest refraction axis.

Here is the Rx Prescribed: O.S. -4.50D / -1.75D x 80°

If vision is acceptable, perform a slit lamp examination to assess adequate fit (centration and movement). If fit is acceptable, dispense the lenses instructing the patient to return in one week for reassessment (see dispensing and follow-up information in PATIENT MANAGEMENT).

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

#### MONOVISION FITTING GUIDELINES

#### A. Patient Selection

#### 1. Monovision Needs Assessment

For a good prognosis, the patient should have adequately corrected distance and near visual acuity in each eye. The amblyopic patient or the patient with significant astigmatism (greater than 1.00D) in one eye may not be a good candidate for monovision correction with these lenses.

Occupational and environmental visual demands should be considered. If the patient requires critical vision (visual acuity and stereopsis), it should be determined by trial whether this patient can function adequately with monovision correction. Monovision contact lens wear may not be optimal for activities such as:

- visually demanding situations such as operating potentially dangerous machinery or performing other potentially hazardous activities; and
- driving automobiles (e.g., driving at night). Patients who cannot meet state driver's licensing requirements with monovision correction should be advised to not drive with this correction, OR may require that additional over-correction be prescribed.

#### 2. Patient Education

All patients do not function equally well with monovision correction. Patients may not perform as well for certain tasks with this correction as they have with spectacles (multifocal, bifocal, trifocal, readers, progressives). Each patient should understand that monovision, as well as other presbyopic alternatives, can create a vision compromise that may reduce visual acuity and depth perception for distance and near tasks. Therefore, caution should be exercised when the patient is wearing the correction for the first time until they are familiar with the vision provided in visually challenging environments (e.g., reading a menu in a dim restaurant, driving at night in rainy/foggy conditions, etc.). During the fitting process, it is necessary for the patient to realize the disadvantages as well as the advantages of clear near vision and straight ahead and upward gaze that monovision contact lenses provide.



#### **B. Eye Selection**

#### 1. Ocular Preference Determination Methods

Generally, the non-dominant eye is corrected for near vision. The following two methods for eye dominance can be used.

- Method 1: Determine which eye is the "sighting eye." Have the patient point to an object at the far end of the room.

  Cover one eye. If the patient is still pointing directly at the object, the eye being used is the dominant (sighting) eye.
- Method 2: Determine which eye will accept the added power with the least reduction in vision. Place a hand-held trial lens equal to the spectacle near ADD in front of one eye and then the other while the distance refractive error correction is in place for both eyes. Determine whether the patient functions best with the near ADD lens over the right or left eye.

#### 2. Other Eye Selection Methods

Other methods include the "Refractive Error Method" and the "Visual Demands Method."

#### Refractive Error Method

For anisometropic correction, it is generally best to fit the more hyperopic (less myopic) eye for distance and the more myopic (less hyperopic) eye for near.

#### Visual Demands Method

Consider the patient's occupation during the eye selection process to determine the critical vision requirements. If a patient's gaze for near tasks is usually in one direction, correct the eye on that side for near.

Example: A secretary who places copy to the left side of the desk will function best with the near lens on the left eye.

## C. Special Fitting Characteristics

#### 1. Unilateral Vision Correction

There are circumstances where only one contact lens is required. As an example, an emmetropic patient would only require a near lens, whereas a bilateral uld require corrective tenses on

both eyes.

#### Examples:

A presbyopic emmetropic patient who requires a +1.75D ADD would have a +1.75D lens on the near eye and the other eye left without correction.

A presbyopic patient requiring a +1.50D ADD who is -2.50D myopic in the right eye and -1.50D myopic in the left eye may have the right eye corrected for distance and the left uncorrected for near.

#### 2. Near ADD Determination

Always prescribe the lens power for the near eye that provides optimal near acuity at the midpoint of the patient's habitual reading distance. However, when more than one power provides optimal reading performance, prescribe the least plus (most minus) of the powers.

#### 3. Trial Lens Fitting

A trial fitting is performed in the office to allow the patient to experience monovision correction. Lenses are fit according to the GENERAL FITTING GUIDELINES for base curve selection described in this Package Insert.

Case history and standard clinical evaluation procedure should be used to determine the prognosis. Determine the distance correction and the near correction. Next determine the near ADD. With trial lenses of the proper power in place, observe the reaction to this mode of correction.

Allow the lenses to settle for about 20 minutes with the correct power lenses in place. Walk across the room and have the patient look at you. Assess the patient's reaction to distance vision under these circumstances. Then have the patient look at familiar near objects such as a watch face or fingernails. Again assess the reaction. As the patient continues to look around the room at both near and distance objects, observe the reactions. Only after these vision tests are completed should the patient be asked to read print. Evaluate the patient's reaction to large print (e.g., typewritten copy) at first and then graduate to newsprint and finally smaller type sizes.

After the patient's performance under the above conditions is correspond tests of and reacting ability runder

conditions of moderately dim illumination should be attempted.

An initial unfavorable response in the office, while indicative of a guarded prognosis, should not immediately rule out a more extensive trial under the usual conditions in which a patient functions.

#### 4. Adaptation

Visually demanding situations should be avoided during the initial wearing period. A patient may at first experience some mild blurred vision, dizziness, headaches, and a feeling of slight imbalance. You should explain the adaptational symptoms to the patient. These symptoms may last for a brief minute or for several weeks. The longer these symptoms persist, the poorer the prognosis for successful adaptation.

To help in the adaptation process, the patient can be advised to first use the lenses in a comfortable familiar environment such as in the home.

Some patients feel that automobile driving performance may not be optimal during the adaptation process. This is particularly true when driving at night. Before driving a motor vehicle, it may be recommended that the patient be a passenger first to make sure that their vision is satisfactory for operating an automobile. During the first several weeks of wear (when adaptation is occurring), it may be advisable for the patient to only drive during optimal driving conditions. After adaptation and success with these activities, the patient should be able to drive under other conditions with caution.

# D. Other Suggestions

The success of the monovision technique may be further improved by having the patient follow the suggestions below:

- Have a third contact lens (distance power) to use when critical distance viewing is needed.
- Have a third contact lens (near power) to use when critical near viewing is needed.
- Having supplemental spectacles to wear over the monovision contact lenses for specific visual tasks may improve the success of monovision correction. This is particularly applicable for those patients who cannot meet state driver's licensing requirements with monovision correction.
- Make use of proper when sarrying out wishal tasks.

Monovision fitting success can be improved by the following suggestions:

- Reverse the distance and near eyes if a patient is having trouble adapting.
- Refine the lens powers if there is trouble with adaptation. Accurate lens power is critical for presbyopic patients.
- Emphasize the benefits of clear near vision and straight ahead and upward gaze with monovision.

The decision to fit a patient with monovision correction is most appropriately left to the Eye Care Professional in conjunction with the patient after carefully considering the patient's needs.

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

#### PATIENT MANAGEMENT

#### **Dispensing Visit**

Each sterile lens is supplied in a foil-sealed plastic package containing buffered saline solution with methyl ether cellulose. To remove the lens from the container, peel back the foil seal, place a finger on the lens, and slide the lens up the side of the bowl of the lens package until it is free of the container.

- Evaluate the physical fit and visual acuity of the lens on each eye.
- Teach the patient how to apply and remove his or her lenses.
- Explain daily disposable lens wear and schedule a follow-up examination.
- Provide the patient with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

REVIEW THESE INSTRUCTIONS WITH THE PATIENT SO THAT HE OR SHE CLEARLY UNDERSTANDS THE PRESCRIBED WEARING AND REPLACEMENT SCHEDULES.

#### **Follow-Up Examinations**

Follow-up care (necessary to ensure continued successful contact lens wear) should include routine periodic progress examinations, management of specific problems, if any, and a proper lens handling procedures.


# Recommended Follow-up Examination Schedule (complications and specific problems should be managed on an individual patient basis):

- 1. One week from the initial lens dispensing to patient
- 2. One month post-dispensing
- 3. Every three to six months thereafter

**NOTE:** Preferably, at the follow-up visits, lenses should be worn for at least six hours.

#### **Recommended Procedures for Follow-up Visits:**

- 1. Solicit and record patient's symptoms, if any.
- 2. Measure visual acuity monocularly and binocularly at distance and near with the contact lenses.
- Perform an over-refraction at distance and near to check for residual refractive error.
- With the biomicroscope, judge the lens fitting characteristics (as described in the **GENERAL FITTING GUIDELINES**) and evaluate the lens surface for deposits and damage.
- 5. Following lens removal, examine the cornea and conjunctiva with the biomicroscope and fluorescein (unless contraindicated).
  - The presence of vertical corneal striae in the posterior central cornea and/or corneal neovascularization is indicative of excessive corneal edema.
  - The presence of corneal staining and/or limbal-conjunctival hyperemia can be indicative of an unclean lens, a reaction to solution preservatives, excessive lens wear and/or a poorly fitting lens.
  - Papillary conjunctival changes may be indicative of an unclean and/or damaged lens.
- Periodically perform keratometry and spectacle refractions. The values should be recorded and compared to the baseline measurements.

If any observations are considered to alleviate the problem and restore the eye to optimal conditions. If


the criteria for successful fit are not satisfied during any follow-up examinations, repeat the patient's trial fitting procedure and refit the patient.

# **WEARING SCHEDULE**

The wearing schedule should be determined by the Eye Care Professional. Regular checkups, as determined by the Eye Care Professional, are also extremely important.

Patients tend to overwear the lenses initially. The Eye Care Professional should emphasize the importance of adhering to the initial maximum wearing schedule. Maximum wearing time should be determined by the Eye Care Professional based upon the patient's physiological eye condition, because individual response to contact lenses varies.

The maximum suggested wearing time for these lenses is:

| Day | Hours |
|-------------|------------------|
| 1 | 6-8 |
| 2 | 8-10 |
| 3 | 10-12 |
| 4 | 12-14 |
| 5 and after | all waking hours |

# REPLACEMENT SCHEDULE

These lenses are indicated for daily disposable wear and should be discarded upon removal.

# LENS CARE DIRECTIONS

When lenses are prescribed for daily disposable wear, the Eye Care Professional should provide the patient with appropriate and adequate warnings and instructions for daily disposable lens wear at the time they are dispensed.


The Eye Care Professional should review with patients that no cleaning or disinfection is needed with daily disposable lenses. Patients should always dispose of lenses when they are removed and have spare lenses or spectacles available.

#### **Basic Instructions**

- Always wash, rinse, and dry hands before handling contact lenses.
- Do not use saliva or anything other than the recommended solutions for lubricating or rewetting lenses. Do not put lenses in the mouth.
- Eye Care Professionals may recommend a lubricating/rewetting solution which can be used to wet (lubricate) lenses while they are being worn to make them more comfortable.

#### Care for a Sticking (Non-Moving) Lens

If the lens sticks (stops moving), the patient should be instructed to apply a few drops of the recommended lubricating or rewetting solution directly to the eye and wait until the lens begins to move freely on the eye before removing it. If non-movement of the lens continues after a few minutes, the patient should immediately consult the Eye Care Professional.

# **EMERGENCIES**

The patient should be informed that if chemicals of any kind (household products, gardening solutions, laboratory chemicals, etc.) are splashed into the eyes, the patient should: FLUSH EYES IMMEDIATELY WITH TAP WATER AND IMMEDIATELY CONTACT THE EYE CARE PROFESSIONAL OR VISIT A HOSPITAL EMERGENCY ROOM WITHOUT DELAY.

# **HOW SUPPLIED**

Each UV-blocking sterile lens is supplied in a foil-sealed plastic package containing buffered saline solution with methyl ether cellulose. The plastic package is marked with the following:

- ACUVUE OASYS® 1-Day: base curve, power, diameter, lot number, and expiration date
- ACUVUE OASYS® 1-Day for ASTIGMATISM: base curve, power, diagnetism, cylinder, axis, and expiration robust that

# REPORTING OF ADVERSE REACTIONS

All serious adverse experiences and adverse reactions observed in patients wearing these lenses or experienced with these lenses should be reported to:

> Johnson & Johnson Vision Care, Inc. 7500 Centurion Parkway Jacksonville, FL 32256 USA

Tel: 1-800-843-2020 www.acuvue.com

JJ

Johnson & Johnson Vision Care, Inc. 7500 Centurion Parkway Jacksonville, FL 32256 USA

Tel: 1-800-843-2020 **www.acuvue.com** 



©Johnson & Johnson Vision Care Companies 2016 In Canada: Johnson & Johnson Vision Care, division of Johnson & Johnson, Inc. In USA: Johnson & Johnson Vision Care, Inc.

Printed in USA. Revision date: 09/16

Revision number: AO-03-16-13



# Clinical Study Protocol Johnson & Johnson Vision Care, Inc.

# LENS FITTING CHARACTERISTICS SUBJECT REPORTED OCULAR SYMPTOMS DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS BIOMICROSCOPY SCALE DISTANCE AND NEAR VISUAL ACUITY EVALUATION TORIC FIT EVALUATION ETDRS DISTANCE VISUAL ACUITY MEASURMENT PROCEDURE PATIENT REPORTED OUTCOMES LENS INSERTION AND REMOVAL VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION

**TESTING**
LENS FITTING CHARACTERISTICS

### SUBJECT REPORTED OCULAR SYMPTOMS

DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS

| Title: | Determination of Distance Spherocylindrical Refractive Error | |
|---|---|---|
| <b>Document Type:</b> | | |
| <b>Document Number:</b> | | <b>Revision Number: 5</b> |
| _ | | |
| _ | | |

BIOMICROSCOPY SCALE













#### DISTANCE AND NEAR VISUAL ACUITY EVALUATION

TORIC FIT EVALUATION



Document Number: Revision Number: 7



**ETDRS DISTANCE VISUAL ACUITY MEASURMENT PROCEDURE** 

Page 1 of 3



Page 3 of 3

### PATIENT REPORTED OUTCOMES

| Title: | Patient Reported Outcomes | | |
|---|---|---|---|
| Document Type: Document Number: | | Revision Number: | 3 |
LENS INSERTION AND REMOVAL

VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION TESTING



APPENDIX F: GUIDELINES FOR COVID-19 RISK MITIGATION

#### 1.0 PURPOSE

The purpose of this document is to provide guidelines for the re-opening or initiation of clinical study sites participating in Johnson & Johnson Vision Care, Inc. (JJVCI) clinical studies during the COVID-19 pandemic.

#### 2.0 SCOPE

This document provides guidelines for Johnson & Johnson Vision Care (JJVCI) to address the potential risks from COVID-19 to study subjects, investigators, study site staff, and monitors at study sites. The guidance provided in this document is in effect from the date of approval through the date of retirement of this Work Instruction. At a minimum, this Work Instruction will be reviewed and updated on a quarterly basis, as appropriate.

NOTE: Re-opening of sites outside of the US will be evaluated on a country by country basis subject to local health authority guidance.

## 3.0 **DEFINITIONS**

American Academy of Optometry (AAO): The American Academy of Optometry is an organization of optometrists based in Orlando, Florida. Its goal is to maintain and enhance excellence in optometric practice, by both promoting research and the dissemination of knowledge. The AAO holds an annual meeting, publishes a monthly scientific journal, gives credentials to optometrists through the fellowship process and publishes position statements.

American Optometric Association (AOA): The American Optometric Association, founded in 1898, is the leading authority on quality care and an advocate for our nation's health, representing more than 44,000 Doctors of Optometry (O.D.), optometric professionals, and optometry students. Doctor of Optometry take a leading role in patient care with respect to eye and vision care, as well as general health and well-being. As primary health care providers, Doctor of Optometry have extensive, ongoing training to examine, diagnose, treat and manage ocular disorders, diseases and injuries and systemic diseases that manifest in the eye. The American Optometric Association is a federation of state, student, and armed forces optometric associations. Through these affiliations, the AOA serves members consisting of optometrists, students of optometry, paraoptometric assistants and technicians. The AOA and its affiliates work to provide the public with quality vision and eye care.

**Centers for Disease Control and Prevention (CDC):** The Centers for Disease Control and Prevention is a national public health institute in the United States. It is a United States federal agency, under the Department of Health and Human Services, and is headquartered in Atlanta, Georgia.

**COVID-19:** Current outbreak of respiratory disease caused by a novel coronavirus. The virus has been named "SARS-CoV-2" and the disease it causes has been named "Coronavirus Disease 2019" (COVID-19).

Clinical Study: Voluntary research studies conducted in people and designed to answer specific questions about the safety or effectiveness of drugs, vaccines, other therapies, or new ways of using existing treatments. May also be called clinical trials, studies, research, trials, or protocols.

Clinical Study Site: Location where a clinical study is conducted, such as a doctor's office, university, or laboratory. Clinical studies are conducted by Investigators who are individual(s) responsible for the conduct of the clinical study at a study site. If a study is conducted by a team of individuals, the Investigator is the responsible leader of the team and may be called the Principal Investigator.

**Clinical Operations Manager (COM):** The Johnson & Johnson Vision Care (JJVCI) individual responsible for the overall management of a clinical trial.

| Title: | Guidelines for CO | Guidelines for COVID-19 Risk Mitigation |
|---|---|---|
| <b>Document Type:</b> | | |
| <b>Document Number:</b> | | Revision Number: 5 |

**Monitor:** An individual designated to oversee the progress of a clinical study and ensure that it is conducted, recorded, and reported in accordance with the protocol, Standard Operating Procedures (SOPs), Good Clinical Practice (GCP), and applicable regulatory requirements.

**Medical Safety Officer (MSO):** Physician who has primary accountability in their product portfolio for product health and safety, and who serves as an independent medical voice for patient safety.

**Safety Management Team (SMT):** A cross-functional, collaborative team responsible for review, assessment and evaluation of medical safety data arising from any source throughout the product life cycle.

#### 4.0 GUIDANCE FOR STUDY DOCUMENTS

In alignment with recent health authority guidance, JJVCI is providing recommendations for study-related management in the event of disruption to the conduct of the clinical study. This guidance does not supersede any local or government requirements or the clinical judgement of the investigator to protect the health, safety and well-being of participants and site staff. If, at any time, a participant's safety is considered to be at risk, study intervention will be discontinued, and study follow-up will be conducted as outlined in the protocol.

During the COVID-19 pandemic, the additional risks listed below need to be considered for study participants and study personnel:

#### 4.1 Additional Risks Related to the COVID-19 Pandemic:

- The possible transmission of the Coronavirus infection and consequent complications, beyond the risk of adverse events due to the investigational device and/or procedures.
- The risk may be higher in an optometric clinical study because of the close contact the subject will have with health care professionals during the procedures and assessments (since the investigator must make the measurements close to the subject's face) and, in addition the need for multiple follow-up visits/exams which may expose the subject to other patients and/or healthcare professionals who might be transmitting the virus, even if they do not have symptoms.
- Potential disruptions to the study may be necessary due to current or future pandemic-related emergency restrictions, which may lead to delays in scheduled follow-up visits.
- Subjects experiencing an adverse event related to contact lens wear may receive delayed treatment
  due to COVID-19 restrictions. In this event, all assessments that can be conducted virtually will be
  completed by the investigator to determine the best course of treatment for the subject, including
  an unscheduled visit, up to discontinuation from the study, as appropriate.

If a study subject is found to have contracted COVID-19 during participation in a study, he/she will be discontinued from the study and followed until COVID-19 Adverse Event (AE) resolution.

To help minimize the above potential risks, JJVCI recommend reviewing/complying with local, state, and governmental guidance for COVID-19 risks.

JJVCI will provide the following study specific documents with language pertaining to COVID-19 risks:

#### 4.1.1 Informed Consent:

Will include information concerning the study-associated risks related to the COVID-19 pandemic in bold font and/or boxed on the first page of the Informed Consent document:

| Title: | Guidelines for COVID-19 Risk Mitigation | 1 |
|---|---|---|
| <b>Document Type:</b> | | |
| <b>Document Number:</b> | | Revision Number: 5 |

#### STUDY ASSOCIATED RISKS RELATED TO COVID-19 (CORONAVIRUS) PANDEMIC

It is important to note that this study will be conducted, at least in part, during the COVID-19 pandemic. As such, additional risks associated with the infection with COVID-19 exist for you. This is particularly important for this study due, in part, to the closeness of the doctor during the study examinations.

The potential effects of the disease are not fully known, at this time, and may include long-term serious health consequences. In severe cases, this may result in hospitalization and/or death. Based on current knowledge from the Centers for Disease Control and Prevention (CDC), those at high-risk for severe illness from COVID-19 include older adults and people with underlying medical conditions.

During this study, all appropriate measures will be taken to minimize risks including the use of personal protective equipment such as masks and gloves, as well as proper sanitization. This is in conformance to guidance from the CDC, local health departments, and the state and county in which the study doctor's office is located. However, these measures may not completely eliminate the risks associated with contracting COVID-19.

If you are found to have contracted COVID-19 or feel ill with flu-like symptoms during participation in the study, you will not be permitted to continue in-office study follow-up visits, but you will receive instructions and your condition will be monitored by the doctor and/or study staff.

#### 4.1.2 COVID-19 Risk Control Checklist (Attachment-B):

Will include COVID-19 risk control methods that are required by a site to conduct JJVCI clinical studies. The risk controls are consistent with CDC, AOA, AAO Guidance. The Principal Investigator will review/sign the study specific checklist prior to the Site Initiation Meeting.

## 4.1.3 Protocol Compliance Investigator(s) Signature Page:

Will include a statement indicating that the Principal Investigator (PI) agrees to conduct the study in compliance with all local, state, and governmental guidance's for COVID-19 risk mitigation.

I have read the suggested guidance provided by JJVCI pertaining to the COVID-19 risk mitigation, (COVID-19 Work Instruction in the Appendix of this protocol). I agree to conduct this study in compliance with local, state, governmental guidance for COVID-19 risks.

## 4.1.4 Study Site Initiation Training Slides:

Will include suggestions to help mitigate potential transmission of COVID-19. Suggestions may include maintaining social distancing in the clinical site by staggered scheduling of study patients, wearing proper PPEs, frequent disinfection, and installing shields on the slit lamp and other applicable equipment.

#### 5.0 GUIDANCE FOR REMOTE SUBJECT VISITS

Potential disruptions to the study may be necessary due to current or future pandemic-related emergency restrictions. Possible disruption of the study as a result of COVID-19 control measures may lead to delays in scheduled follow-up visits.

Subjects may be delayed in being seen for study follow up visit(s), for example due to COVID-19 control measures or due to the subject's concerns or fears about COVID-19 risk. When appropriate, the remote assessment will be conducted to the extent possible. Discussions with the subject during remote assessments may include:

Title:
Document Type:

Document Number: Revision Number: 5

| Procedure | Details |
|---|---|
| Subject Reported Ocular<br>Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire regarding the test article when applicable and feasible. |
| Change of Medical History<br>(Adverse Events) and<br>Concomitant Medications /<br>Therapies Review | Record any adverse events or medical history changes from the previous study visit with the subject/parents. Review the subject's concomitant medications/therapies and record any changes from the previous study visit. |
| Wearing Time and Compliance | any changes from the previous study visit. Record the average wearing time (including number of hours per day during weekdays and weekends, and number of days per week). Confirm compliance with the prescribed wear schedule. Record and discuss the lens wear compliance based on the subject's self-report. For example, the subjects will be asked the time of the day the subject typically puts on the study lenses in the morning and takes off in the evening, the number of days per week lenses were worn, and the number of consecutive days the subject didn't wear the study lenses, etc. |

The discussion with the subject will be documented in EDC under Tele-Visit and a minor protocol deviation will be noted. If during the telephone consultation, a subject states he/she wishes to discontinue participating in the study, instruct the subject to stop wearing the study lenses and schedule the subject to return to the clinic for a Final Evaluation at the at earliest possible time. Subjects should return all unused lenses to the clinic at the last visit.

Changes in study visit schedules, missed visits, or participant discontinuations may lead to missing data, including data related to protocol-specified procedures. Case report forms should capture specific information regarding the basis of missing data, including the relationship to the COVID-19 pandemic.

#### 6.0 STUDY CONDUCT DURING PANDEMIC

It is recognized that the Coronavirus Disease 2019 (COVID-19) pandemic may have an impact on the conduct of this clinical study due to, for example, self-isolation/quarantine by participants and study-site personnel; travel restrictions/limited access to public places, including Optometry Clinics; and changes in clinic procedures required to address the COVID-19 challenge.

Every effort should be made to adhere to protocol-specified assessments for study participants, including follow-up. However, if scheduled visits cannot be conducted in person at the study site it is suggested that assessments be performed to the extent possible remotely/virtually or delayed until such time that on-site visits can be resumed in order to continue participant monitoring in accordance with the protocol where possible. At each contact, participants will be interviewed to collect safety data. Key efficacy endpoint assessments should be performed if required and as feasible.

Modifications to protocol-required assessments may be permitted via COVID-19 Appendix after consultation with the participant, investigator, and the sponsor. Missed assessments/visits will be captured in the clinical trial management system for protocol deviations. Interruptions of test article wear or discontinuations of study interventions and withdrawal from the study should be documented with the prefix "COVID-19-related" in the case report form (CRF).

| Title: | Guidelines for CO | DVID-19 Risk Mitigation |
|-------------------------|-------------------|-------------------------|
| <b>Document Type:</b> | | |
| <b>Document Number:</b> | | Revision Number: 5 |

The sponsor will continue to monitor the conduct and progress of the clinical study, and any changes will be communicated to the sites and to the health authorities according to local guidance.

If a participant has tested positive for COVID-19, the investigator should contact the sponsor's responsible medical monitor to discuss initial plans for study intervention and follow-up. The medical monitor will notify the Safety Management Team of any subject(s) that have reported "COVID-19", "Asymptomatic COVID-19", or "Suspected COVID-19" adverse events within 24 hours of the notification.

Modifications made to the study conduct as a result of the COVID-19 pandemic will be summarized in the clinical study report.

COVID-19 screening procedures that may be mandated by local healthcare systems do not need to be reported as an amendment to the protocol even if done during clinical study visits.

### 6.1 Monitoring Visits

When on-site monitoring by the sponsor is not feasible, the sponsor's site monitor will contact the study site to schedule remote visits. In such cases, on-site monitoring visits will resume when feasible, with increased frequency to address the source data verification backlog.

Even with staffing limitations during this COVID-19 pandemic, all routine operations related to clinical trials should be well-documented and archived as part of standard process. When conditions permit, all parties involved in this clinical trial should communicate relevant information in a timely manner so that all relevant parties remain sufficiently informed.

### 6.1.1 Study Site Initiation:

During the period that this Work Instruction is in effect, Site Initiation Meetings and training of study site staff will be conducted remotely. The JJVCI study team will conduct training via Skype, Zoom, Microsoft Teams or similar software as well as utilize online training materials, as applicable. Study site training will be documented utilizing Site Initiation Report per Study Site Initiation

On-site visits may be considered when, for example, hands-on training or evaluation of site facilities is required. While on site, the Clinical Research Associate (CRA) will follow all local, state, and governmental policies for COVID-19 Risk Mitigation, including social distancing, wearing of PPE, etc. as applicable for the location of the study site.

## 6.1.2 Interim Monitoring Visits (if applicable):

During the period that this Work Instruction is in effect, Interim Monitoring On-site visits will be kept to a minimum and include only those tasks that the CRA cannot perform remotely (e.g., source document verification, test article reconciliation, etc.).

To ensure data integrity during the conduct of all JJVC studies, clinical study teams will follow the study specific Clinical Monitoring Plan

While on site, the CRA will follow all local, state, and governmental policies for COVID-19 Risk Mitigation, including social distancing, wearing of PPE, etc. as applicable for the location of the study site.

| Title: | <b>Guidelines for COVID-19 Risk Mitigation</b> | |
|---|---|---|
| <b>Document Type:</b> | | |
| <b>Document Number:</b> | | Revision Number: 5 |

# 6.1.3 Study Site Closure:

During the period that this Work Instruction is in effect, the duration of the Study Site Closure Visit will be limited to tasks that the CRA cannot perform remotely (e.g., source document verification, test article final reconciliation and return, etc.).

| Title: | Guidelines for COVID-19 Risk Mitiga | tion |
|---|---|---|
| <b>Document Type:</b> | | |
| <b>Document Number:</b> | | Revision Number: 5 |

### **Attachment A: Study Site Correspondence**

XXXX XX, 2020

## Re: COVID-19 Mitigation Plan, <<CR-xxxx/protocol title>>

Dear << Principal Investigator>> and Study Team,

Coronavirus (COVID-19) has impacted several communities and business activities over the past several months. While we work toward the successful conduct of clinical studies, our commitment continues to be the safety of patients, healthcare professionals, and to our communities.

Therefore, we would like to share the following revisions/additions related to the above referenced Johnson & Johnson Vision Care company sponsored clinical trial(s) you are currently working on or considering participation within.

#### **Protocol:**

• Guidelines for COVID-19 Risk Mitigation provided in the Appendix section.

#### **Protocol Signature Page:**

 Will include a statement indicating the Principal Investigator agrees to conduct the study in compliance with all local, state, and governmental guidelines for COVID-19 risk mitigation.

## **Informed Consent:**

• Will include information concerning the study-associated risks related to the COVID-19 pandemic in bold font and/or boxed on the first page of the Informed consent document.

## **COVID-19 Risk Control Checklist for Clinical Studies:**

• Will include COVID-19 risk control measures that are required to ensure the safety and health of subjects, site staff and monitors during the pandemic.

We want to encourage the need for open lines of communication about potential challenges you may foresee as the result of the current COVID-19 situation. Therefore, we encourage you to regularly connect with your respective Johnson & Johnson clinical study team (Clinical Research Associate (CRA), Lead CRA or Study Managers).

Thank you for your continued engagement, collaboration, and dedication to your study subjects during this challenging time.

Please file this letter in your site file study correspondence.

| Title: | Guidelines for COVID-19 Risk Mitigation | 1 |
|---|---|---|
| <b>Document Type:</b> | | |
| <b>Document Number:</b> | | Revision Number: 5 |

# **COVID-19 Risk Control Checklist (Attachment-B):**

Study Number Site Number Principal Investigator (PI) Name

The following COVID-19 risk control methods are required to conduct Johnson & Johnson Vison Care clinical studies. Please review the following requirements and Initial each requirement.

| PI Initials | General Site Safety Planning Measures |
|---|---|
| | Signage within site describing Risk Control methods |
| | Social Distancing practices throughout site (waiting rooms, lobby, exam rooms, etc.) |
| | Non-contact thermometer available to assess temperatures of staff and patients |
| | Training on patient flow and physical distancing in waiting room |
| | Establish longer time frame between patient appointments to reduce persons in the site |
| | Staff should receive job-specific training on PPE and demonstrate competency with selection and proper use of PPE and wear at all times during interactions with subjects (e.g., putting on and removing without self-contamination) |

| PI Initials | Site Staff Daily Safety Measures |
|---|---|
| | As part of routine practice, site staff should regularly monitor themselves for fever and symptoms |
| | of COVID-19, including temperature checks |
| | Any staff member (including non-study clinic staff and Investigators) showing signs of being sick |
| | or testing positive for COVID-19 must not be permitted to work on activity that may expose study |
| | related staff and subject and the Sponsor shall be informed |
| | NOTE: Inform JJVC in 24 hours of any COVID-19 cases and all potential exposure during |
| | the clinical study. |
| | Ensure that all staff wear a mask |
| | Gloves should be required when working directly with patients and changed between each patient |
| | Have staff thoroughly wash hands for at least 20 seconds or use an alcohol-based hand sanitizer |
| | when they arrive, before and after each patient, before eating and after using the bathroom. |
| | Cleaning and disinfection procedures for exam rooms and instruments or equipment between |
| | patients with gloves. |
| | Cleaning and disinfection procedures for commonly touched surfaces (doors, chairs, computers, |
| | phones, etc.) with gloves. |

| PI Initials | Before a Patient or Study Visit: |
|---|---|
| | Patients should be asked prior to entering the site about fever and respiratory illness and whether they or a family member have had contact with another person with confirmed COVID-19 in the past 14 days. Patients exhibiting signs of being sick should be rescheduled when their symptoms resolve. |
| | Instruct patients that companions should remain outside of the facility and not accompany the patient into the facility unless they are a parent/guardian of the patient or if they are a true caregiver and need to assist the patient |
| | Request the patient to call or text the office upon arrival so entrance to and movement through facility can be coordinated by site staff |

| Title: | Guidelines for COVID-19 Risk Mitigation | 1 |
|---|---|---|
| <b>Document Type:</b> | | |
| <b>Document Number:</b> | | Revision Number: 5 |

| PI Initials | Patients Entering the site: |
|---|---|
| | Temperature checks utilizing a non-contact thermometer for all patients and companions entering |
| | the site. |
| | All patients and companions must wear cloth or disposable mask at all times in the site |
| | Maintain social distancing. Waiting rooms or lobbies should be as empty as possible. Advise |
| | seated patients to remain at least 6 feet from one another. |
| | Communal objects in (e.g. toys, reading materials, etc.) should be removed or cleaned regularly. |

I certify that I have read and agree to implement all the listed COVID-19 Risk Control Measures required for the conduct of Johnson & Johnson Vision Care studies.

Principal Investigator Signature and Date

| Title: | Guidelines for CC | Guidelines for COVID-19 Risk Mitigation | |
|---|---|---|---|
| <b>Document Type:</b> | | | |
| Document Number | | , | Revision Number: 5 |

## **RESOURCE LINKS**

#### **US Resource Links**

OSHA Training

https://www.osha.gov/SLTC/covid-19/controlprevention.html

Personal Protective Equipment (PPE) Training

CDC: https://www.cdc.gov/coronavirus/2019-ncov/hcp/using-ppe.html

I&R Training

ACUVUE® LensAssist: https://www.acuvue.com/lensassist

• Clinic Preparedness Guides

CDC: <a href="https://www.cdc.gov/coronavirus/2019-ncov/hcp/clinic-preparedness.html">https://www.cdc.gov/coronavirus/2019-ncov/hcp/clinic-preparedness.html</a>
AOA: <a href="https://aoa.uberflip.com/i/1240437-aoa-guidance-for-re-opening-practices-covid-19/1?m4="https://www.aoa.org/optometry-practice-reactivation-preparedness-guide">https://www.aoa.org/optometry-practice-reactivation-preparedness-guide</a>

• In-Office Disinfection of Multi-Patient Use Diagnostic Contact Lenses

<a href="https://www.gpli.info/wp-content/uploads/2020/03/2020-01-15-in-office-disinfecting-of-diagnostic-lenses.pdf">https://www.gpli.info/wp-content/uploads/2020/03/2020-01-15-in-office-disinfecting-of-diagnostic-lenses.pdf</a>

#### **OUS Resource Links**

- Updates on local regulations in Hong Kong https://www.coronavirus.gov.hk/eng/index.html
- Resumption of optical services in England: Letter from Matt Neligan and Poonam Sharma <a href="https://www.england.nhs.uk/coronavirus/wp-content/uploads/sites/52/2020/04/C0601-reopening-of-optical-services-letter-17-june-2020.pdf">https://www.england.nhs.uk/coronavirus/wp-content/uploads/sites/52/2020/04/C0601-reopening-of-optical-services-letter-17-june-2020.pdf</a>
- NHS Optical Letter
   <a href="https://www.england.nhs.uk/coronavirus/wp-content/uploads/sites/52/2020/04/C0127-optical-letter-1-april-2020.pdf">https://www.england.nhs.uk/coronavirus/wp-content/uploads/sites/52/2020/04/C0127-optical-letter-1-april-2020.pdf</a>
- The College of Optometrists primary eye care COVID-19 guidance: Red phase
   https://www.college-optometrists.org/the-college/media-hub/news-listing/coronavirus-covid-19-guidance-for-optometrists.html
- The College of Optometrists COVID-19: College updates https://www.college-optometrists.org/the-college/media-hub/news-listing/coronavirus-2019-advice-for-optometrists.html#CollegeGuidelines
- Infection Control Guidelines. (n.d.). Retrieved from Canadian Association Of Optometrists: https://opto.ca/sites/default/files/resources/documents/infection\_control\_guidelines\_2016.pdf
- Infection prevention and control for COVID-19: Interim guidance for outpatient and ambulatory care settings. (2020, May 23 May). Retrieved from Government of Canada: https://www.canada.ca/en/public-health/services/diseases/2019-novel-coronavirus-infection/guidance-documents/interim-guidance-outpatient-ambulatory-care-settings.html

| Title: | <b>Guidelines for COVID-19 Risk Mitigation</b> | |
|---|---|---|
| <b>Document Type:</b> | | |
| <b>Document Number:</b> | | <b>Revision Number: 5</b> |

- Information for Members On Coronavirus (COVID-19). (n.d.). Retrieved from Canadian Association Of Optometrists:
  - $https://opto.ca/sites/default/files/resources/documents/information\_for\_members\_on\_coronavirus.pdf$
- Coronavirus (COVID-19) resources for health professionals, including aged care providers, pathology providers and health care managers. (2020, September 24). Retrieved from Australian Government Department of Health:
  - https://www.health.gov.au/resources/collections/coronavirus-covid-19-resources-for-health-professionals-including-aged-care-providers-pathology-providers-and-health-care-managers
- Environmental Cleaning and Disinfection Principles for COVID-19. (n.d.). Retrieved from Australian Government Department of Health: https://www.health.gov.au/sites/default/files/documents/2020/03/environmental-cleaning-and-disinfection-principles-for-covid-19.pdf
- Infection control guidelines and advice. (n.d.). Retrieved from Optometry Australia: https://www.optometry.org.au/practice-professional-support/coronavirus-covid-19-what-optometrists-need-to-know/covid-19-clinical-advice/infection-control-guidelines-and-advice/

## PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE

Protocol Number and Title: CR-6484 Evaluation of Toric Soft Contact Lenses Containing a Chromophore to Block High-Energy Visible Light Produced on Commercial Manufacturing Lines

Version and Date: 1.0 14 March 2022

I have read and understand the protocol specified above and agree on its content.

I agree to conduct this study according to ISO 14155:2020,<sup>1</sup> GCP and ICH guidelines,<sup>2</sup> the Declaration of Helsinki,<sup>3</sup> United States (US) Code of Federal Regulations (CFR),<sup>4</sup> and the pertinent individual country laws/regulations and to comply with its obligations, subject to ethical and safety considerations. The Principal Investigator is responsible for ensuring that all clinical site personnel, including Sub-Investigators adhere to all ICH<sup>2</sup> regulations and GCP guidelines regarding clinical trials during and after study completion.

I will assure that no deviation from or changes to the protocol will take place without prior agreement from the Sponsor and documented approval from the Institutional Review Board (IRB), except where necessary to eliminate an immediate hazard(s) to the trial participants.

I am responsible for ensuring that all clinical site personnel including Sub-Investigators adhere to all ICH<sup>2</sup> regulations and GCP guidelines regarding clinical trials during and after study completion.

All clinical site personnel involved in the conduct of this study have completed Human Subjects Protection Training.

I agree to ensure that all clinical site personnel involved in the conduct of this study are informed about their obligations in meeting the above commitments.

I shall not disclose the information contained in this protocol or any results obtained from this study without written authorization.

I have read the suggested guidance provided by JJVCI pertaining to the COVID-19 risk mitigation, (COVID-19 Work Instruction in Appendix F of this protocol). I agree to conduct this study in compliance with local, state, governmental guidance for COVID-19 risks.

| Principal<br>Investigator: | | |
|----------------------------|------------------------------------------|------|
| | Signature | Date |
| Institution/Site: | Name and Professional Position (Printed) | |
| | Institution/Site Name | |
| | Institution/Site Address | |